Replication of the PARADIGM-HF Heart Failure Trial in Healthcare Claims Data

DUPLICATE PARADIGM-HF January 25, 2021

NCT04736433

#### 1. RCT Details

This section provides a high-level overview of an RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Angiotensin-Neprilysin Inhibition versus Enalapril in Heart Failure (PARADIGM-HF trial)

#### 1.2 <u>Intended aim(s)</u>

The primary objective of the study is to determine LCZ696 200 mg twice daily, a combination of sacubitril/valsartan, is superior to enalapril 10 mg twice daily in reducing the composite endpoint in place of Angiotensin Converting Enzyme inhibitors (ACEi) and Angiotensin II receptor blockers (ARBs)

#### 1.3 Primary endpoint for replication and RCT finding

Composite endpoint of death from cardiovascular (CV) causes or hospitalization for heart failure (HF)

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

After following 8000 patients for 34 months, at an overall two-sided alpha level of 0.05, the primary end point would occur in 2410 patients, which would provide a power of 97% to detect a 15% reduction in the risk of this outcome.

#### 1.5 Trial estimate

HR = 0.80 (95% CI 0.73–0.87) comparing LCZ696 to enalapril (McMurry et al., 2014, NEJM)

#### 2. Person responsible for implementation of replication in Aetion

Helen Tesfaye, Pharm.D, ScM implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of design and analytic choices. All implementation steps are recorded, and implementation history is archived in the platform.

#### 3. Data Source(s)

Optum Cliniformatics Data Mart, IBM MarketScan, Medicare

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expediated review

#### Design Diagram - PARADIGM-HF TRIAL REPLICATION



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group retrospective cohort study design comparing sacubitril/valsartan to ACE inhibitors. Although the trial compared sacubitril/valsartan to enalapril, we expanded the definition of the comparator group to include all ACEi therapies to improve power, since all medications within this class of medication are indicated and guideline recommended for use in heart failure with reduced ejection fraction patients and would be expected to have similar effects on the primary outcome of CV death and HF hospitalization.

The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of sacubitril/valsartan or a ACEi (cohort entry).

#### 5.2 Important steps for cohort formation

New users (defined as no use of sacubitril/valsartan in 180 days prior to index date) of the exposure will be identified. New users of a comparator drug were identified as patients with no ACEi fills during the 60 days prior to the index date to allow for patients who are switching among ACEi drugs or restarting ACEi after a brief lapse.

#### 5.2.1 Eligible cohort entry date

Sacubitril/valsartan was approved by FDA for market availability on July 7, 2015.

- Optum: July 7, 2015 March 31, 2020 (end of data availability)
- Marketscan: July 7, 2015 December 31, 2018 (end of data availability)
- Medicare: July 7, 2015 December 31, 2017 (end of data availability)

#### 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

| | Opt | um | Marke | etscan | Medi | care* |
|---|---|---|---|---|---|---|
| | Less Excluded | Remaining | Less Excluded | Remaining | Less Excluded | Remaining |
| | Patients | Patients | Patients | Patients | Patients | Patients |
| All patients | | 77,673,639 | | 200,203,908 | | 23,466,175 |
| Did not meet cohort entry criteria | -73,445,846 | 4,227,793 | -196,533,760 | 3,670,148 | -18,348,713 | 5,117,462 |
| Excluded due to insufficient enrollment | -623,954 | 3,603,839 | -340,051 | 3,330,097 | -1,288,867 | 3,828,595 |
| Excluded due to prior use of referent | -3,168,921 | 434,918 | -2,967,886 | 362,211 | -3,495,789 | 332,806 |
| Excluded due to prior use of exposure | -29,778 | 405,140 | -12,511 | 349,700 | -33,013 | 299,793 |
| Excluded because patient qualified in >1 exposure category | -8 | 405,132 | -3 | 349,697 | -9 | 299,784 |
| Excluded based on Age | 0 | 405,132 | -1 | 349,696 | 0 | 299,784 |
| Excluded based on Gender | -39 | 405,093 | 0 | 349,696 | 0 | 299,784 |
| Excluded based on Inclusion #1 - Age >=18 years old | -624 | 404,469 | -1,354 | 348,342 | -721 | 299,063 |
| Inclusion #3 - HFrEF prediction algorithm applied to reference group† | -381,531 | 22,938 | -337,242 | 11,100 | -259,816 | 39,247 |
| Excluded based on Inclusion #4b - Hospitalization for HF within the last 12 months | -9,321 | 13,617 | -4,618 | 6,482 | -10,685 | 28,562 |
| Excluded based on Inclusion #5a - ACEis or ARBs | -1,224 | 12,393 | -385 | 6,097 | -1,534 | 27,028 |
| Excluded based on Inclusion #5b - Beta-blockers | -673 | 11,720 | -248 | 5,849 | -2,128 | 24,900 |
| Excluded based on Exclusion #3 - Known history of angioedema | -56 | 11,664 | -29 | 5,820 | -200 | 24,700 |
| Excluded based on Exclusion #4 - Treatment with both ACEis AND ARBs | -15 | 11,649 | -9 | 5,811 | -34 | 24,666 |
| Excluded based on Exclusion #5 - Acute decompensated HF | -1,060 | 10,589 | -435 | 5,376 | -5,457 | 19,209 |
| Excluded based on Exclusion #6 - Symptomatic hypotension | -734 | 9,855 | -240 | 5,136 | -1,964 | 17,245 |
| Excluded based on Exclusion #7 - Low eGFR / renal dysfunction | -1,064 | 8,791 | -403 | 4,733 | -2,833 | 14,412 |
| Excluded based on Exclusion #8 - Hyperkalemia | -57 | 8,734 | -14 | 4,719 | -116 | 14,296 |
| Excluded based on Exclusion #9 - ACS, Stroke, TIA, CABG, PCI, Other CV Procedures, Carotid Angioplasty | -765 | 7,969 | -546 | 4,173 | -2,912 | 11,384 |
| Excluded based on Exclusion #11 - Implantation of CRT device | -41 | 7,928 | -19 | 4,154 | -1,550 | 9,834 |
| Excluded based on Exclusion #12 - History of heart transplant or LVAD | -56 | 7,872 | -33 | 4,121 | -35 | 9,799 |
| Excluded based on Exclusion #13 - History of severe pulmonary disease | -463 | 7,409 | -205 | 3,916 | -1,029 | 8,770 |
| Excluded based on Exclusion #14 - Diagnosis of peripartum-<br>or chemotherapy-induced cardiomyopathy | -38 | 7,371 | -34 | 3,882 | -60 | 8,710 |

| Excluded based on Exclusion #15 - Documented untreated ventricular arrhythmia with syncopal episodes | -18 | 7,353 | -6 | 3,876 | -25 | 8,685 |
|---|---|---|---|---|---|---|
| Excluded based on Exclusion #16 - Second- and third-degree AV block | -73 | 7,280 | -29 | 3,847 | -73 | 8,612 |
| Excluded based on Exclusion #17 - Presence of haemodynamically significant mitral and/or aortic valve disease | -124 | 7,156 | -43 | 3,804 | -246 | 8,366 |
| Excluded based on Exclusion #19a - History of active inflammatory bowel disease (IBD) | -18 | 7,138 | -12 | 3,792 | -37 | 8,329 |
| Excluded based on Exclusion #19b - Active duodenal/gastric ulcers | -13 | 7,125 | -8 | 3,784 | -25 | 8,304 |
| Excluded based on Exclusion #19c - Evidence of hepatic disease | -173 | 6,952 | -80 | 3,704 | -265 | 8,039 |
| Excluded based on Exclusion #19d - Current treatment with cholestyramine or colestipol resins | 0 | 6,952 | 0 | 3,704 | -4 | 8,035 |
| Excluded based on Exclusion #21 - Ivabradine use | -6 | 6,946 | -10 | 3,694 | -4 | 8,031 |
| Final cohort | | 6,946 | | 3,694 | | 8,031 |

<sup>\*</sup> The Medicare data cut included all patients with a diagnosis for HF, stroke, or diabetes.

#### 6 Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of sacubitril/valsartan (ARNi) at any dose and frequency. Initiation will be defined by no use of sacubitril/valsartan during the prior 180 days before treatment initiation (washout period). Patients are required to be incident users with respect to their exposure group only, since one of the RCT inclusion criteria was prior treatment with ACEi or ARB.

#### **Comparator agents:**

Initiators of ACEi, any dose and frequency.

#### 6.2 <u>Preliminary Covariates:</u>

Age

<sup>†</sup> Algorithm provided in Desai et al. (2018).

- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period of 180 days prior to and including the index prescription date

Covariates listed above are a small subset of covariates that will ultimately be controlled in the design and analysis phase of the study. They are included in the preliminary assessment to determine the presence of adequate overlap between the two population of patients to proceed to the next phase of the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and initial power assessment and are listed in Table 1 (Appendix B).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Composite of hospitalization for heart failure and all-cause mortality
- Secondary outcomes:
  - Heart failure hospitalization
  - o All-cause death

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted, definitions provided in Appendix A):

1. Bleeding (we expect to see a null association, as renin angiotensin aldosterone inhibitors are not expected to have any impact on this outcome)

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analysis will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analysis, the follow-up will start the day after the initiation of sacubitril/valsartan or ACEi and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continue registration in the database,
- End of the study period,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (sacubitril/valsartan or ACEi) + a 30-day grace period,
- The date of switching from an exposure to comparator and vice versa,
- The date of switching to or initiation of any angiotensin II receptor blockers (ARBs), including combination medications containing ARBs,
- The date of switching to or initiation of aliskiren, including combination therapies.

For the ITT analyses, the censoring based on the switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7 Initial Feasibility Analysis

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/1069/results/61863/result/0
Marketscan- https://bwh-dope.aetion.com/projects/details/1072/results/61852/result/0

Medicare - https://bwh-dope.aetion.com/projects/details/1073/results/61854/result/0

#### Date conducted: 11/24/2020

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome.

- Complete study flowchart from Section 5.3
- Report patient characteristics by treatment group

| Optum | Marketscan | Medicare |
|-------|------------|--------------|
| | | 111001100110 |

| Variable | Reference -<br>ACE inhibitors | Exposure -<br>Sacubitril/valsa<br>rtan | Difference | Reference -<br>ACE inhibitors | Exposure -<br>Sacubitril/valsa<br>rtan | Difference | Reference -<br>ACE Inhibitors | Exposure -<br>Sacubitril/valsa<br>rtan Copy | Differ |
|---|---|---|---|---|---|---|---|---|---|
| Number of patients | 4,217 | 2,729 | - | 2,218 | 1,476 | - | 6,293 | 1,738 | _ |
| Age | 1 | | 1 | | ' | | | ' | |
| mean (sd) | 66.94 (13.39) | 68.39 (12.07) | -1.45 (-2.06, -<br>0.84) | 60.86 (14.92) | 61.21 (13.50) | -0.36 (-1.29 <i>,</i><br>0.57) | 77.16 (8.29) | 76.04 (7.56) | 1.12 (<br>1.5 |
| median<br>[IQR] | 68.00 [58.00,<br>77.00] | 70.00 [61.00,<br>77.00] | - | 60.00 [52.00,<br>71.00] | 60.00 [53.00,<br>70.00] | - | 76.00 [70.00,<br>84.00] | 75.00 [70.00,<br>81.00] | |
| Gender | <br> | | <br> | | | | | | <u> </u> |
| Males; n (%) | 2,829 (67.1%) | 1,773 (65.0%) | 2.1% (-0.2%,<br>4.4%) | 1,606 (72.4%) | 1,018 (69.0%) | 3.4% (0.4%,<br>6.5%) | 3,433 (54.6%) | 1,003 (57.7%) | -3.2% (-<br>0.5 |
| Females; n<br>(%) | 1,388 (32.9%) | 956 (35.0%) | -2.1% (-4.4%,<br>0.2%) | 612 (27.6%) | 458 (31.0%) | -3.4% (-6.5%, -<br>0.4%) | 2,860 (45.4%) | 735 (42.3%) | 3.2% (<br>5.8 |
| CCI (180 days)-<br>ICD9 and<br>ICD10 v2 | | | | | | | | | |
| mean (sd) | 6.52 (2.50) | 6.70 (2.24) | -0.18 (-0.29, -<br>0.06) | 5.51 (2.22) | 5.70 (2.04) | -0.19 (-0.33, -<br>0.05) | 7.53 (2.91) | 7.00 (2.51) | 0.53 (<br>0.6 |
| median<br>[IQR] | 6.00 [5.00,<br>8.00] | 6.00 [5.00,<br>8.00] | - | 5.00 [4.00,<br>7.00] | 5.00 [4.00,<br>7.00] | - | 7.00 [5.00,<br>9.00] | 7.00 [5.00,<br>9.00] | - |

### Report summary parameters of study population

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Variable | Value | Value | Value |
| Number of patients in full cohort | 6,946 | 3,694 | 8,031 |
| Number of patients dropped as incomplete cases | 0 | 0 | 2 |
| Number of patients that did not begin follow-up | 16 | 5 | 7 |
| Number of patients in analytic cohort | 6,930 | 3,689 | 8,022 |

| Number of events | 1435 | 592 | 1992 |
|---|---|---|---|
| Number of person-years | 3,277.04 | 1,877.04 | 3,093.20 |
| Number of patients in group: ACE Inhibitors - Reference | 4,208 | 2,216 | 6,286 |
| Number of patients in group: Sacubitril/Valsartan - Exposure | 2,722 | 1,473 | 1,736 |
| Risk per 1,000 patients | 207.07 | 160.48 | 248.32 |
| Rate per 1,000 person-years | 437.9 | 315.39 | 643.99 |

Report median follow-up time by treatment group

| Patient Group | Optum<br>Median Follow-Up<br>Time (Days) [IQR] | Marketscan<br>Median Follow-Up<br>Time (Days) [IQR] | Medicare<br>Median Follow-Up<br>Time (Days) [IQR] |
|---|---|---|---|
| Overall Patient Population | 95 [43, 213] | 117 [58, 242] | 82 [39, 173] |
| Referent - ACE Inhibitors | 99 [42, 209] | 118 [58, 240] | 81 [38, 170] |
| Exposure - Sacubitril/Valsartan | 92 [44, 217] | 111 [57, 246] | 86 [45, 183] |

• Report reasons for censoring in the overall study population

| | Optum | Marketscan | Medicare |
|---|---|---|---|
| Overall | 6930 | 3689 | 8022 |
| Outcome | 1,361 (19.6%) | 558 (15.1%) | 1,933 (24.1%) |
| Start of an additional exposure | 252 (3.6%) | 155 (4.2%) | 156 (1.9%) |
| End of Index Exposure | 2,445 (35.3%) | 1,264 (34.3%) | 2,078 (25.9%) |
| Specified date reached | 1,101 (15.9%) | 721 (19.5%) | 1,964 (24.5%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 645 (9.3%) | 713 (19.3%) | 691 (8.6%) |
| Switch to ARBs or Aliskiren + Nursing Home admission Occurred | 1,126 (16.2%) | 278 (7.5%) | 1,200 (15.0%) |

#### 8 Initial Power Assessment

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1069/results/61862/result/0">https://bwh-dope.aetion.com/projects/details/1069/results/61862/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1072/results/61853/result/0">https://bwh-dope.aetion.com/projects/details/1072/results/61853/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1073/results/61855/result/0">https://bwh-dope.aetion.com/projects/details/1073/results/61855/result/0</a>

Date conducted: 11/24/2020

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index.

• In the appropriate excel sheet below, report number of patients matched in each treatment group. Input the overall risk of outcome from Section 7. Input the desired or assumed HR, alpha level, and non-inferiority margin (if applicable) from the RCT (Section 1.3.1). The number of expected events and corresponding power are then calculated automatically. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together.

| , | Onture | Marketscan | Medicare | Pooled |
|---|---|---|---|---|
| | Optum | iviarketscan | iviedicare | Pooled |
| Number of people matched | | | | |
| Reference | 2722.0 | 1468.0 | 1736.0 | 5926.0 |
| Exposure | 2722.0 | 1468.0 | 1736.0 | 5926.0 |
| Risk per 1,000 patients | 207.1 | 160.5 | 248.3 | |
| Rate per 1,000 person-years | 437.9 | 315.4 | 644.0 | |
| N of events | 1,435 | 592 | 1,992 | 4,019 |
| N of patients (both groups) at Step 1 | | | | |
| in or patients (both groups) at step 1 | 6,946 | 3,694 | 8,031 | 18,671 |
| Risk per 1,000 patients | 206.6 | 160.3 | 248.0 | 215.3 |

| Superiority Analysis (Pooled) | |
|-------------------------------|------------|
| Number of patients matched | |
| Reference | 5,926 |
| Exposed | 5,926 |
| Risk per 1,000 patients | 215.25 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 2551.143 |
| Power | 0.99988126 |

| Superiority Analysis (Optum) | |
|------------------------------|-----------|
| Number of patients matched | |
| Reference | 2,722 |
| Exposed | 2,722 |
| Risk per 1,000 patients | 207.10 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1127.4524 |
| Power | 0.9629782 |

| Superiority Analysis (Marketscan) | |
|-----------------------------------|-------------|
| Number of patients matched | |
| Reference | 1,468 |
| Exposed | 1,468 |
| Risk per 1,000 patients | 160.50 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 471.228 |
| Power | 0.677969637 |

| Superiority Analysis (Medicare) | |
|---------------------------------|-------------|
| Number of patients matched | |
| Reference | 1,736 |
| Exposed | 1,736 |
| Risk per 1,000 patients | 248.30 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 862.0976 |
| Power | 0.905904762 |

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/2/20 |
|---|---|---|---|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 12/8/20 |
| Reasons for stopping analysis (if required): | | | |

#### 9. Balance Assessment

Optum- <a href="https://bwh-dope.aetion.com/projects/details/1069/results/63131/result/0">https://bwh-dope.aetion.com/projects/details/1069/results/63131/result/0</a>
Marketscan- <a href="https://bwh-dope.aetion.com/projects/details/1073/results/63128/result/0">https://bwh-dope.aetion.com/projects/details/1073/results/63128/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/1073/results/63128/result/0">https://bwh-dope.aetion.com/projects/details/1069/results/63129/result/0</a>

Date conducted: 12/22/2020

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the

dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

• Report covariate balance after matching.

Note- For Table 1, please refer to **Appendix B**.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0%) | 0 (0%) | 0 (0%) |
| Death | 150 (2.47%) | 64 (2.11%) | 86 (2.84%) |
| Start of an additional exposure | 309 (5.09%) | 106 (3.49%) | 203 (6.69%) |
| End of Index Exposure | 2285<br>(37.67%) | 1206<br>(39.76%) | 1079<br>(35.58%) |
| Specified date reached | 1868 (30.79) | 879<br>(28.98%) | 989<br>(32.61%) |
| End of patient enrollment | 696<br>(11.47%) | 366<br>(12.07%) | 330<br>(10.88%) |
| Switch to ARBs or<br>Aliskiren + Nursing<br>Home admission<br>Occurred | 758<br>(12.50%) | 412<br>(13.58%) | 346<br>(11.41%) |

• Report follow-up time by treatment group.

| Patient Group | Optum<br>Median<br>Follow-Up Time<br>(Days) [IQR] | Marketscan<br>Median<br>Follow-Up Time<br>(Days) [IQR] | Medicare<br>Median<br>Follow-Up Time<br>(Days) [IQR] |
|---|---|---|---|
| Overall Patient Population | 118 [58, 286] | 139 [59, 296] | 102 [46, 189] |
| Referent - ACE Inhibitors | 126 [60, 309] | 142 [77, 295] | 102 [42, 170] |
| Exposure - Sacubitril/Valsartan | 108 [56, 266] | 136 [58, 300] | 106 [58, 218] |

• Report overall risk of the primary outcome.

| | Optum | MarketScan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 206.6 | 160.3 | 248.0 | 215.3 |

#### 6. Final Power Assessment

Date conducted: 12/22/2020

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

| Superiority Analysis (Pooled) | |
|-------------------------------|-------------|
| Number of patients matched | |
| Reference | 3,033 |
| Exposed | 3,033 |
| Risk per 1,000 patients | 215.25 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1305.7065 |
| Power | 0.980850168 |

| 1,279 |
|-------------|
| 1,279 |
| 206.60 |
| 0.8 |
| 0.05 |
| 528.4828 |
| 0.727390963 |

| Superiority Analysis (Marketscan) | |
|-----------------------------------|-------------|
| Number of patients matched | |
| Reference | 748 |
| Exposed | 748 |
| Risk per 1,000 patients | 160.30 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 239.8088 |
| Power | 0.408308308 |

| Superiority Analysis (Medicare) | |
|---------------------------------|-------------|
| Number of patients matched | |
| Reference | 1,006 |
| Exposed | 1,006 |
| Risk per 1,000 patients | 248.30 |
| Desired HR from RCT | 0.8 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 499.5796 |
| Power | 0.703266933 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 12/26/20 |
|-------------------------|------------------|----------------|----------|
| Reviewed by FDA: | | Date reviewed: | |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### References

Desai RJ, Lin KJ, Patorno E, et al. Development and Preliminary Validation of a Medicare Claims—Based Model to Predict Left Ventricular Ejection Fraction Class in Patients With Heart Failure. Circ: Cardiovascular Quality and Outcomes. 2018;11(12). doi:10.1161/CIRCOUTCOMES.118.004700

McMurray JJV, Packer M, Desai AS, et al. Angiotensin–Neprilysin Inhibition versus Enalapril in Heart Failure. New England Journal of Medicine. 2014;371(11):993-1004. doi:10.1056/NEJMoa1409077

| # | PARADIGM-HF trial definitions | Implementation in routine care | Please see the following Google Drive for further details or<br>https://drive.google.com/drive/folders/1WD618wrywYjE. | |
|---|---|---|---|---|
| | Trial details - active comparision - 2 wee | ICD-10 codes are not listed in this document because of excel cell size lim 10 codes. Full ICD-10 code lists will be available in the above Google Drix code conversions were completed using a SAS macro that implements for CMS ICD-9 to ICD-10 mapping: https://www.nber.org/data/icd9-icd- equivalence-mapping.html | ve Folder (link above). ICD-9 to ICD-10 ward/ backward mapping based on the | |
| | EXPOSURE vs. COMPARISON | V | References/Rationale | Color coding |
| | LCZ696 (sacubitril/valsartan) 200 mg twice daily vs. enalapril 10 mg twice daily | Sacubitril/valsartan vs. enalapril | | |
| | Aim: To determine if LCZ696 is superior to enalapril in reducing the risk of death and of hospitalization for HF | Exposure: new-use of sacubitril/valsartan Reference: enalapril | | |
| | PRIMARY OUTCOME | <u>Exposure</u> : new-use of sacobitn/valsartan <u>Reference</u> , enalapin | | Criteria Adequate mapping in claims |
| | The primary outcome is a composite of death from cardiovasclar causes or hositalization for heart failure | Measured 14 days after drug initiation in diagnosis position specified below and inpatient care setting: Hospital admission for CHF (Inpatient only, any position) ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 ICD-10 diagnosis: 150.1, 150.2x, 150.4, 150.814, 109.81, 111.0 (hypertensive heart disease with HF), 113.0 | | Intermediate mapping in claims |
| | INCLUSION CRITERIA | | | Poor mapping or cannot be measure in claims |
| 1 | Age ≥ 18 years | Age 18 years or older at drug initiation | | Can't be measured in claims but not<br>important for the analysis |
| 2 | NYHA functional class II–IV | Measured 45 days prior to and including the day of <u>oral</u> drug initiation in generic prescription claims requiring 28 days supply of Loop or Thiazide diuretics Loop Diuretics: Burnetanide, Furosemide, Torsemide, Ethacrynic acid -OR- Thiazide and Thiazide-like Diuretics: Hydrochiorothiazide, Chlorothiazide, Chlorthalidone, Indapamine, Metolazone, Cyclothiazide, Hydroflumethiazide, Benzthiazide, Methyclothiazide, Polythiazide | | |
| 3 | LVEF ≤ 35% | Measured 180 days prior to and including the day of index drug initiation in any diagnosis position and inpatient or outpatient care setting Systolic Heart Failure ICD-9 diagnosis: 428.2x ICD-10 diagnosis: 150.2x Combined Systolic/Diastolic Heart Failure ICD-9 diagnosis: 428.4x ICD-10 diagnosis: 150.4x | | |
| 4 | Plasma BNP≥150 pg/mL or NT-proBNP≥600 pg/mL at the screening visit and a hospitalization for HF within the last 12 months | | | |
| 4a | Plasma BNP ≥150 pg/mL or NT-proBNP ≥600 pg/mL at the screening visit | | | |
| ı | AND the following: | | | J |

| | The company of the co | |
|---|---|---|
| Hospitalization for heart failure within the last 12 months | Meaured 365 days prior to drug initiation in any diagnosis position and inpatient care setting Hospital Admission for CHF. ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 ICD-10 diagnosis: I50.1, I50.2x, I50.4, I50.814, I09.81, I11.0, I13.0, I13.2 | |
| Treatment with a <b>stable dose</b> of an ACE inhibitor <b>or</b> an ARB <b>equivalent</b> to <b>enalapril 10 mg/day</b> for at least 4 weeks before the screening visit; and treatment with a stable dose of a beta-blocker for at least 4 weeks prior to the screening visit, unless contraindicted or not tolerated | | |
| Treatment with a <b>stable dose</b> of an ACE inhibitor <b>or</b> an ARB <b>equivalent to enalapril 10 mg/day</b> for at least <b>4</b> weeks before the screening visit | Measured 47 days to 2 days prior to drug initiation in prescription claims requiring 28 days supply of oral ACE inibitors' generic names for prescription claims: Enalapril, Captopril, Cilazapril, Fosinopril, Lisinopril, Moexipril, Perindopril, Quinapril, Ramipril, Trandolapril, Zofenopril, Benazepril -OR- ARBs generic names for prescription claims: Candesartan, Eprosartan, Irbesartan, Losartan, Olmesartan, Telmisartan, Valsartan, Azilsartan | |
| AND the following. | Magazinal 45 days prior to index drug initiation in processing claims (generic names) of an oral | |
| Treatment with a <b>stable dose of a beta-blocker for at least 4 weeks</b> prior to the screening visit, unless contraindicated or not tolerated | beta-blocker for at least 4 weeks (28 days) Beta-blocker generic names for prescription claims: | |
| Although not required, the protocol specified that an aldosterone antagonist should also be considered in all patients, taking account of renal function, serum potassium, and tolerability. If given, the dose of aldosterone antagonist should be stable for at least 4 weeks prior to the screening visit | | |
| EXCLUSION CRITERIA | | |
| History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACE inhibitors (ACEIs), ARBs, or neprilysin inhibitors, as well as known or suspected contraindications to the study drugs | | |
| Previous history of intolerance to recommended target doses of ACEIs or ARBs | | |
| Known history of angioedema | Measured from the start of all available data to index drug initiation in any diagnosis position and inpatient or outpatient care setting ICD-9 diagnosis: 995.1 ICD-10 diagnosis: 778.3x | |
| Requirement for treatment with <b>both ACEIs and ARBs</b> | Measured 180 days prior to and including day of drug initiation in prescription claims (generic names) for any of oral ACE initiators (generic names) for any of oral ACE initiators (generic names for prescription claims: Enalapril, Captopril, Cilazapril, Fosinopril, Lisinopril, Moexipril, Perindopril, Quinapril, Ramipril, Trandolapril, Zofenopril, Benazepril -AND- ARBs generic names for prescription claims: Candesartan, Eprosartan, Irbesartan, Losartan, Olmesartan, Telmisartan, Valsartan, Azilsartan | |
| Current acute decompensated heart failure (exacerbation of chronic heart failure manifested by signs and symptoms that may require intravenous therapy) | Measured 7 days prior to and including day of drug initiation in any diagnosis position and inpatient and emergency care setting ICD-9 diagnosis: 428.41, 428.43 ICD-10 diagnosis: I50.23, I50.41, I50.43 | |
| Symptomatic hypotension and/or a systolic blood pressure <100 mmHg at Visit 1 (screening) or <95 mmHg at Visit 3 or at Visit 5 (randomization) | Measured 30 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Hypotension: ICD-9 diagnosis: 458.xx, 785.5x ICD-10 diagnosis: 195.xx, R57.xx | |
| | Treatment with a stable dose of an ACE inhibitor or an ARB equivalent to enalapril 10 mg/day for at least 4 weeks before the screening visit; and treatment with a stable dose of a beta-blocker for at least 4 weeks prior to the screening visit, unless contraindicted or not tolerated Treatment with a stable dose of an ACE inhibitor or an ARB equivalent to enalapril 10 mg/day for at least 4 weeks before the screening visit Treatment with a stable dose of an ACE inhibitor or an ARB equivalent to enalapril 10 mg/day for at least 4 weeks before the screening visit AND the following: Treatment with a stable dose of a beta-blocker for at least 4 weeks prior to the screening visit, unless contraindicated or not tolerated Although not required, the protocol specified that an aldosterone antagonist should also be considered in all patients, taking account of renal function, serum potassium, and tolerability. If given, the dose of aldosterone antagonist should be stable for at least 4 weeks prior to the screening visit EXCLUSION CRITERIA History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACE inhibitors (ACEIs), ARBs, or neprilysin inhibitors, as well as known or suspected contraindications to the study drugs Previous history of intolerance to recommended target doses of ACEIs or ARBs Known history of angloedema Requirement for treatment with both ACEIs and ARBs Current acute decompensated heart failure (exacerbation of chronic heart failure manifested by signs and symptoms that may require intravenous therapy) Symptomatic hypotension and/or a systolic blood pressure <100 mmHg at Visit 1 (screening) or <35 mmHg at Visit 3 or at | So de algorison College Colleg |

| | | Measured 30 days prior to and including day of drug initiation in any diagnosis position and inpatient |
|---|---|---|
| | | or outpatient care setting |
| | | Acute kidney injury (AKI). ICD-9 diagnosis: S84:xx, 586 |
| | | ICD-10 diagnosis: 584.xx, 586<br>ICD-10 diagnosis: N17.x, N19 |
| | | Acute glomerulnephritis |
| | | ICD-9 diagnosis: S80.xx<br>ICD-10 diagnosis: N00.3, N00.8, N00.9, N01.3 |
| | Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 at Visit 1 (screening), Visit 3 (end of enalapril run-in), or | Chronic Kidney Disease (CKD) - Stage IV and V |
| 7 | Visit 5 (end of LCZ696 run-in and randomization) or >35% decline in eGFR between Visit 1 and Visit 3 or between Visit 1 and | ICD-9 diagnosis: 585.4, 585.5<br>ICD-10 diagnosis: N18.4, N18.5 |
| | Visit 5 | ESRD |
| | | ICD-9 diagnosis: 403.01, 403.11, 403.91, 404.03, 404.13, 585.6 |
| | | ICD-10 diagnosis: I12.0, N18.6 |
| | | Hemodialysis/Peritoneal Dialysis ICD-9 diagnosis: V45.1x, V56.xx, 996.56, 996.68, 996.73 |
| | | ICD-10 diagnosis: Z49.xx, Z91.15, Z99.2, T85.611x, T85.621x, T85.631x, T85.691x, T85.71x<br>ICD-9 procedure: 39.95, 54.98 |
| | | ICD-10 procedure: 5A1D70Z, 5A1D80Z, 5A1D90Z, 3E1M39Z<br>CPT-4 code: 90935, 90937, 90939 |
| | | Measured 30 days prior to and including day of drug initiation in any diagnosis position and inpatient |
| | | or outpatient care setting |
| 8 | Serum potassium >5.2 mmol/L at Visit 1 (screening) or >5.4 mmol/L at Visit 3 or Visit 5 (randomization) | Hyperkalemia ICD-9 diagnosis: 276.7 |
| | | ICD-10 diagnosis: E87.5 |
| | | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting |
| | | Acute Coronary Syndrome: STEMI & NSTEMI |
| | | ICD-9 diagnosis: 410.xx (exclude 410.x2), 411.0<br>ICD-10 diagnosis: I21.xx, I22.xx, I23.xx |
| | | Acute Coronary Syndrome: Unstable Angina |
| | | ICD-9 diagnosis: 413.xx (exclude 413.1), 411.1, 411.8, 411.81, 411.89<br>ICD-10 diagnosis: I20.xx (exclude I20.1), I24.xx (exclude 124.1) |
| | | Stroke |
| 9 | Acute coronary syndrome, stroke, transient ischaemic attack, cardiac, carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within the 3 months prior to Visit 1. | ICD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.xx ( <i>excluding</i> 434.x0), 436.x, 997.02<br>ICD-10 diagnosis: G97.3x, I60.xx, I61.xx I62.xx, I63.xx, I67.89, I97.81x, I97.82x |
| | | TIA |
| 1 | | ICD-9 diagnosis: 435.xx<br>ICD-10 diagnosis: G45.xx |
| | | CABG/ Transmyocardial Revascularization |
| | | ICD-9 diagnosis: V45.81, 996.03 ICD-10 diagnosis: 295.1 |
| 1 | | ICD-9 procedure: 36.1x, 36.2, 36.3x |
| | | ICD-10 procedure: Refer to "CABG & Revascularization" tab within this spreadsheet for complete list of procedure codes |
| 10 | Coronary or carotid artery disease likely to require surgical or <b>percutaneous intervention within the 6 months after Visit 1</b> | Included above |
| | | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting |
| | | Pacemaker and Implantable cardiac Defibillators: |
| 11 | Implantation of a cardiac resynchronization therapy (CRT) device within 3 months prior Visit 1 or intent to implant a CRT | ICD-9 diagnosis: V45.01, V45.02, V45.09, V53.31, V53.32, 996.01, 996.04, 996.61 ICD-10 diagnosis: Z95.0, 295.810, Z45.010, Z45.018, Z45.02, T82.110A, T82.111A, T82.120A, |
| | | T82.121A, T82.190A, T82.191A, T82.6XXA, T82.7XXA ICD-9 procedure: 00.50, 00.51, 00.53, 00.54, 37.7x, 37.8x, 37.94 - 37.98 |
| | | ICD-10 procedure: Refer to "CRT_Implant" tab CPT-4 code: 33200 - 33208, 33220 - 33229, 33230 - 33238, 33240 - 33249, 33262 - 33264, 33270, |
| | | 33271, 93640 - 93642, 93280 - 93289, 93290 - 93299 |

| | | | 1 |
|---|---|---|---|
| 12 | | Measured from all available data to and including the day of drug initiation in any diagnosis position and inpatient or outpatient care setting Heart Transplantation ICD-9 diagnosis: V42.1, V49.83, 996.83 ICD-10 diagnosis: 294.1, 276.82, 786.20, 786.21, 786.22 ICD-9 procedure: 33.6, 37.51 ICD-10 procedure: 33.6, 37.51 ICD-10 procedure: 02YA0Z0, 02YA0Z1, 02YA0Z2 CPT-4 code: 33935, 33945 LVAD/Implantable Heart ICD-9 diagnosis: V43.2x ICD-10 diagnosis: 295.811, 295.812 ICD-9 procedure: 37.60, 37.66 ICD-10 procedure: 02HA0RS, 02HA3RS, 02HA4RS, 5A02116, 5A02216, 02HA0QZ, 02HA3QZ, 02HA4QZ CPT-4 code: 33975, 33976, 33979, 33981 - 33983, 33977, 33978, 33980 | |
| 13 | History of severe pulmonary disease | Measured from all available data to and including day of drug initiation in any diagnosis position and in inpatient or outpatient care setting Worsening Asthma/Status Asthmaticus ICD-9 diagnosis: 493.01, 493.02, 493.11, 493.12, 493.2x, 493.91, 493.22 ICD-10 diagnosis: 145.21, 145.22, 145.901, 145.902 COPD/Chronic Tuberclosis ICD-9 diagnosis: 491.xx, 492.xx, 494.x, 496, 506.4, 748.61, 011.5x ICD-10 diagnosis: 141.x, 143.x, 147.x, 144.x, 168.4, Q33.4, A15.0 Pulmonary Firbrosis or Interstitial Lung Disease (ILD) ICD-9 diagnosis: 515.516.3x, 516.8, 516.9 ICD-10 diagnosis: 184.10, 184.111, 184.112, 184.113, 184.114, 184.115, 184.116, 184.117, 184.09, 184.2, 184.89, 184.9 Cystic Fibrosis ICD-9 diagnosis: 277.0x ICD-10 diagnosis: E84.xx Pulmonary Hypertension/Other Pulmonary Heart Disease ICD-9 diagnosis: 127.xx Sarcoldosis | Pulmonary firbrosis/Interstitial lung disease: Jones N, Schneider G, Kachroo S, et al. A systematic review of validated methods for identifying pulmonary fibrosis and interstitial lung disease using administrative and claims data. Pharmacoepidemiol Drug Saf. 2012;21(1):256-60. Available at: http://www.ncbi.nlm.nih.gov/pubmed/22262614. |
| | Diagnosis of peripartum- or chemotherapy-induced cardiomyopathy within the 12 months prior to Visit 1 | Measured from 365 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Peripartum Cardiomyopathy ICD-9 diagnosis: 674.5x ICD-10 diagnosis: 090.3 Chemotherapy-Induced Cardiomyopathy ICD-9 diagnosis: 425.9 ICD-10 diagnosis: 142.7 | |
| | Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months prior to Visit 1 Documented ventricular arrhythmia within the 3 months prior to Visit 1 | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient and outpatient care setting ICD-9 diagnosis: 427.1, 427.4x, 427.5 ICD-10 diagnosis: 147.2, 149.01, 149.02, 146.9 | |
| | AND the following: | | |
| 15 | Syncopal episodes within the 3 months prior to Visit 1 | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient and outpatient care setting Syncopal Episodes ICD-9 diagnosis: 780.2 ICD-10 diagnosis: R55 | |
| 1 | AND the following: | | |

| 150 | Untreated ventricular arrhythmia within the 3 months prior to visit 1 | Measured 90 days prior to and including day of drug initiation WITHOUT any of these non-drug treatments for ventricular tachycardia in any diagnosis position and inpatient and outpatient care setting Implantable Cardioverter-Defbrillator ICD-9 diagnosis: V45.00, V45.02, V45.09, V53.32, 996.04, 996.61 ICD-10 diagnosis: 295.9, 295.810, 295.818, 245.02, T82.110A, T82.111A, T82.120A, T82.121A, T82.190A, T82.191A ICD-9 procedure: 00.51, 00.54, 37.94 - 37.98 ICD-10 procedure: 02HK0KZ, 02HK3KZ, 02HK4KZ, 02HL0KZ, 02HL3KZ, 02HL4KZ, 01H609Z, 01H639Z, 01H839Z O1H809Z, 01H839Z CPT-4 code: 33220, 33223, 33230, 33231, 33240 - 33249, 33262 - 33264, 33270, 93640 - 93642, 93280 - 93285, 93285, 93289, 93292, 93295 | |
|---|---|---|---|
| | OR the following: | | |
| 150 | Untreated ventricular arrhythmia within the 3 months prior to visit 1 | Measured 90 days prior to and including day of drug initiation WITHOUT any of these oral drug treatments for ventricular arrythmia in prescription claims Beta-blockers: Acebutolol, Atenolol, Betaxolol, Bisoprolol, Carteolol, Carvedilol, Labetalol, Metoprolol, Metiranolol, Nebivolol, Nadolol, Propranolol, Pindolol, Sotalol, Penbutolol, Oxprenolol Non-DHP.CCB: Diltiazem, Verapamil Antiarrhythmic drugs: Amiodarone, Procainamide, Mexiletine, Flecainide, Moricizine | |
| 16 | Symptomatic bradycardia or second- or third-degree atrioventricular block without a pacemaker | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient and outpatient care setting | |
| | | Second- and Third-degree AV block<br>ICD-9 diagnosis: 426.0, 426.1x (except 426.11)<br>ICD-10 diagnosis: 144.2, 144.30, 144.1 | |
| 17 | Presence of haemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to LV dilatation | Measured 180 days prior to and including day of drug initiation in any diagnosis position and in inpatient and outpatient care setting ICD-9 diagnosis: 394.0, 395.0, 395.2, 396.0, 396.2, V42.2, V43.3 ICD-10 diagnosis: 105.0, 106.0, 106.2, 108.0, 295.3, 295.2 ICD-9 procedure: 55.01, 35.02, 35.05, 35.06, 35.11, 35.12, 35.21, 35.22, 35.23, 35.24, 35.97 ICD-10 procedure: 02NF3ZZ, 02NF4ZZ, 02NG3ZZ, 02NG4ZZ, 02RF3ZZ, 02RF3ZZ, 02RF3Z, 02RG3Z, 02RG3 | |
| 18 | Presence of other haemodynamically significant obstructive lesions of the LV outflow tract, including aortic and subaortic | Included in the definition of exclusion criterion # 17 | |
| | stenosis | models in the definition of exclusion effection # 17 | |
| 19 | Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study | | |
| 19a | drugs, including, but not limited to, any of the following: History of active inflammatory bowel disease during the 12 months before Visit 1 | Measured 365 days prior to and including day of drug initiation in any diagnosis position in inpatient and outpaient care setting <u>Ulcerative Colitis</u> ICD-9 diagnosis: S56.xx ICD-10 diagnosis: K51.xx <u>Crohn's Disease</u> ICD-9 diagnosis: S55.x ICD-10 diagnosis: K50.xx | Thirumurthi S, Chowdhury R, Richardson P, Abraham NS. Validation of ICD-<br>9-CM diagnostic codes for inflammatory bowel disease among veterans.<br>Dig Dis Sci. 2010 Sep;55(9):2592-8. doi: 10.1007/s10620-009-1074-z. Epub<br>2009 Dec 24. PubMed PMID: 20033847 |
| | OR the following: | | |
| 191 | Active duodenal or gastric ulcers during the 3 months prior to Visit 1 | Measured 90 days prior to and including day of drug initiation in any diagnosis position in inpatient and outpaient care setting <u>Duodenal Ulcers</u> ICD-9 diagnosis: 532.0x, 532.1x, 532.2x, 532.3x, 532.9x ICD-10 diagnosis: k25.0 - k25.3, K25.9 <u>Gastric Ulcers</u> ICD-9 diagnosis: 531.0x, 531.1x, 531.2x, 531.3x, 531.9x ICD-10 diagnosis: K26.0 - K26.3, K26.9 | |
| 1 | OR the following: | | |
| 1 | OR the following: | I | |

| 1 | | Measured from the start of all available data of drug initiation in any diagnosis position in inpatient |
|---|---|---|
| | | and outpaient care setting |
| | | and outpaient care setting |
| | | Hepatic Encephalopathy/Coma |
| | | ICD-9 diagnosis: 070.0, 070.2x, 070.4x, 070.6, 070.71, 572.2 |
| | | ICD-10 diagnosis: B15.0, B16.0, B16.2, B17.11, B19.0, B19.11, B19.21, K72.90, K72.91 |
| | | 100 20 diagnosis. 013:0, 010:0, 010:1, 017:11, 013:0, 013:11, 013:11, 17:130, 17:131 |
| | | Esophageal Varicies |
| | | ICD-9 diagnosis: 456.0, 456.1, 456.2x, 572.3 |
| | | ICD-10 diagnosis: I85.xx, K76.6 |
| | Evidence of hepatic disease as determined by any one of the following: aspartate aminotransferase or alanine | Porto-Caval Shunt |
| 190 | aminotransferase values exceeding 2× upper limit of normal at Visit 1, history of hepatic encephalopathy, history of | ICD-9 procedure: 39.1, 42.91 |
| | oesophageal varices, or history of porto-caval shunt | ICD-10 procedure: Codes are in the sheet 'PCShunt' |
| | | CPT-4 code: 37182, 37183, 37241 |
| | | er i i fer i i i i i e |
| | | <u>Cirrohosis/Chronic Hepatic Diseases</u><br>ICD-9 diagnosis: 571.0, 571.2, 571.3, 571.4, 571.5, 571.6 |
| | | ICD-10 diagnosis: K70.0, K70.30, K70.9, K73.0, K73.2, K73.8, K73.9, K75.4, K74.0, K74.60, K74.69, |
| | | K74.3, K74.4, K74.5, K74.1 |
| | | K/4.3, K/4.4, K/4.3, K/4.1 |
| | | NASH |
| | | ICD-9 diagnosis: 571.8, |
| | | ICD-10 diagnosis; K76.0 |
| | OR the following: | |
| | | Measured 30 days prior to and including the day of index drug initiation for <u>oral</u> generic prescription |
| 19d | Current treatment with cholestyramine or colestipol resins | claims of |
| 130 | | |
| <u> </u> | | Cholestyramine, Colestipol, Colesevelam |
| 20 | Presence of any other disease with a life expectancy of 5 years | Charlson Comborbidity Index > 10 |
| Ľ | The control of the co | and an analysis and an analysi |
| | | Measure since 2015/all available data in drug prescription claims for any dispensings of |
| 21 | Any Ivabradine use Approved in April 2015 (same year as Entresto) | Consideration and the base of the control of the co |
| | | Generic name: Ivabradine Brand name: Corlanor |
| | | Dranu name. Conanor |

| | Variable | Codes and Medications (all medical claims, inpatient and outpatient should be used to define the coniditions unless otherwise specified) | | When Measured for replicating | When Measured<br>(Rishi's algorithm) |
|---|---|---|---|---|---|
| 1 | Intercept | N/A | -1.37219 | | |
| 2 | Cardiomyopathy | ICD-9 diagnosis: 425.x<br>ICD-10 diagnosis: I42.x, I43.x | | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 3 | Diastolic heart failure | ICD-9 diagnosis: 428.3x (not co-occuring with 428.2x ) ICD-10 diagnosis: I50.3x (not co-occuring with I50.2x) | | Measured between 180 days prior to and including the date of drug initiation and pick claim closest to the index initiation | on index date |
| 4 | Left heart failure | ICD-9 diagnosis: 428.1x (not co-occuring with more specific systolic or diastolic HF codes of 428.2x or 428.3x ) ICD-10 diagnosis: I50.1 (not co-occuring with more specific systolic or diastolic HF codes of I50.2x or I50.3x ) | | Measured between 180 days prior to and including the date of drug initiation and pick claim closest to the index initiation | on index date |
| 5 | Systolic heart failure | ICD-9 diagnosis: 428.2x (not co-occuring with 428.3x) ICD-10 diagnosis: I50.2x (not co-occuring with I50.3x) | 0.754954 | Measured between 180 days prior to and including the date of drug initiation and pick claim closest to the index initiation | on index date |
| 6 | Myocardial infarction | ICD-9 diagnosis: 410.xx<br> ICD-10 diagnosis: | | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 7 | Unspecified heart failure | ICD-9 diagnosis: 428.0x, 428.4x, 428.9x, 428.2x PLUS 428.3x<br>ICD-10 diagnosis: I50.4x, I50.8x, I50.9, I50.2x PLUS I50.3x | | Measured between 180 days<br>prior to and including the date<br>of drug initiation and pick claim<br>closest to the index initiation | on index date |
| 8 | Number of hospitalizations for CHF | ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 ICD-10 diagnosis: I50.1, I50.2x, I50.4, I50.814, I09.81, I11.0, I13.0, I13.2 | 0.346289 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date<br>(including index<br>date) |
| 9 | Male gender | Male | 0.323651 | Measured on the date of index drug initiation | on index date |
| 10 | Implantable cardioverter defibrillator | I <u>CD-9 diagnosis</u> : V45.02 I <u>CD-10 diagnosis</u> : Z95.810 I <u>CD-9 procedure</u> : 37.94 - 37.98 I <u>CD-10 procedure</u> : Please copy from ICD-10 codes tabs for implantable cardioverter defibrillator | 0.275032 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |

| 11 | ACE inhibitor | Prescription claims for: Benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril | 0.221748 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
|---|---|---|---|---|---|
| 12 | Index diagnosis recorded during an outpatient visit | Any diagnosis position in an <b>outpatient care setting</b> <u>ICD-9 diagnosis:</u> 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 <u>ICD-10 diagnosis</u> : I50.1, I50.2x, I50.4x, I50.814, I09.81, I11.0, I13.0, I13.2 | -0.187191 | Measured between 180 days prior to and including the date of drug initiation and pick claim closest to the index initiation | on index date |
| 13 | Mineralocorticoid receptor antagonist | <u>Prescription claims for</u> : Eplerenone, spironolactone | 0.166008 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 14 | Anemia | ICD-9 diagnosis: 280.xx - 285.xx ICD-10 diagnosis: Please copy from ICD-10 codes tabs for anemia | -0.165353 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 15 | Valve disorder | ICD-9 diagnosis: 394.x - 397.x, 398.9x, V42.2, V43.3 ICD-10 diagnosis: Please copy from ICD-10 codes tabs for valve disorder ICD-9 procedure: 35.1x, 35.2x ICD-10 procedure: Please copy from ICD-10 codes tabs for valve disorder CPT code: 33660-33665, 33400-33403, 33420-33430, 33460, 33463-33468, 33475, 33496, 0257T, 0258T, 0259T, 0262T | -0.163684 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 16 | Digoxin | <u>Prescription claims for</u> : Digoxin | 0.163224 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 17 | Thiazide diuretic | <u>Prescription claims for</u> : Bendroflumethiazide, Benzthiazide, Chlorothiazide,<br>Chlorthalidone, Hydrochlorothiazide, Indapamide, Methyclothiazide, Metolazone,<br>Polythiazide, Quinethazone, Trichlormethiazide | -0.160819 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 18 | Obesity | ICD-9 diagnosis: 278.00, 278.01, V85.3x, V85.4x ICD-10 diagnosis: E65.x, E66.x, E67.x, E68.x CPT codes: 43842, 43843, 43846, 43847, 43848, G0447 Prescriptions claims for: orlistat, sibutramine, phentermine, benzphetamine, phendimetrazine, diethylpropion | -0.141956 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 19 | Nitrate | <u>Prescription claims for</u> : Nitroglycerin, isosorbide dinitrate, isosorbide mononitrate, ranolazine | 0.129225 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 20 | Other dysrythmias | ICD-9 diagnosis: 427.0x, 427.1x, 427.2x, 427.4x, 427.6x, 427.8x, 427.9x, 785.0x ICD-10 diagnosis: Please copy from ICD-10 tab for other dysrythmias | 0.116652 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 21 | Hypertension | ICD-9 diagnosis: 401.xx, 402.xx, 405.xx<br> ICD-10 diagnosis: 110, 111.0, 111.9, 112.0, 112.9, 113.0, 113.10, 113.11, 113.2, 115.0, 115.1, 115.2, 115.8, 115.9 | -0.098539 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |

| 22 | Beta blocker | Prescription claims for oral: Acebutolol, atenolol, betaxolol, bisoprolol, carteolol, carvedilol, labetalol, metoprolol, nadolol, nebivolol, penbutolol, pindolol, propranolol | 0.087257 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
|---|---|---|---|---|---|
| 23 | Loop diuretic | Prescription claims for oral: Bumetanide, furosemide, torsemide, ethacrynic acid | 0.084251 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 24 | Rheumatic heart disease | <u>ICD-9 diagnosis</u> : 393 - 398.x<br><u>ICD-10 diagnosis</u> : I05.xx - I09.xx | -0.073889 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 25 | Psychosis | ICD-9 diagnosis: 290.8x, 290.9x, 295.xx, 297.xx, 298.xx, 299.xx, 780.0x - 780.5x ICD-10 diagnosis: Please copy from ICD-10 tab for Psychosis | -0.068198 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 26 | Coronary artery bypass graft | <u>ICD-9 procedure</u> : 36.1x, 36.2x<br><u>ICD-10 procedure</u> : Please copy from ICD-10 tab for CABG<br><u>CPT code</u> : 33510 – 33536, 33545, 33572 | -0.040175 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 27 | COPD | ICD-9 diagnosis: 491.xx, 492.xx, 496.xx, 493.2x<br>ICD-10 diagnosis: J41.x, J42.x, J43.x, J44.x | -0.037023 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 28 | Sleep apnea | ICD-9 diagnosis: 327.2x, 780.51, 780.53, 780.57<br>ICD-10 diagnosis: G47.3x | -0.03556 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 29 | Hypertensive nephropathy | ICD-9 diagnosis: 403.xx, 404.xx<br>ICD-10 diagnosis: I12.x, I13.xx | -0.03383 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 30 | Depression | ICD-9 diagnosis: 293.83, 296.2x, 296.3x, 296.9x, 298.0x, 300.4x, 309.1x, 309.28, 311.xx ICD-10 diagnosis: F06.3x, F32.x, F33.x, F34.x, F39.x, F43.21, F43.23 | -0.033829 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 31 | Hypotension | <u>ICD-9 diagnosis</u> : 458.xx<br><u>ICD-10 diagnosis</u> : 195.x | -0.017282 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 32 | Stable angina | ICD-9 diagnosis: 413.xx ICD-10 diagnosis: Please copy from ICD-10 tab for stable angina | -0.015657 | Measured 180 days prior to and including the date of index drug initiation | 6 months prior to<br>index date + index<br>date + 30days post-<br>index |
| 33 | Age | Continous | -0.005747 | Measured on the date of index drug initiation | on index date |

| 34 | Atrial fibrillation | ICD-9 diagnosis: 427.3x<br>ICD-10 diagnosis: I48.x | | Measured 180 days prior to and including the date of index drug initiation | |
|---|---|---|---|---|---|
| 35 | Hyperlipidemia | ICD-9 diagnosis: 272.xx<br>ICD-10 diagnosis: E78.xx | -0.001805 | Measured 180 days prior to and including the date of index drug initiation | inday data + inday |

#### Mortality-Dependent on data source.

1. All-cause mortality / inpatient mortality Identified using the vital status file-

#### Medicare

Identified using the discharge status codes-

#### Optum-

- 20 = EXPIRED
- 21 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 22 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 23 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 24 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 25 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 26 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 27 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 28 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 29 = EXPIRED TO BE DEFINED AT STATE LEVEL
- 40 = EXPIRED AT HOME (HOSPICE)
- 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE)
- 42 = EXPIRED PLACE UNKNOWN (HOSPICE)

#### Truven-

- 20 Died
- 22 Died
- 23 Died
- 24 Died
- 25 Died
- 26 Died
- 27 Died
- 28 Died
- 29 Died
- 40 Other died status or Expired at home (Hospice claims only) (depends on year)
- 41 Other died status or Expired in medical facility (Hospice claims only) (depends on year)
- 42 Other died status or Expired place unknown (Hospice claims only) (depends on year)
- 21 Died or Disch./Transf. to court/law enforcement (depends on year)

| CPT-4 Code Range |
|------------------|
| 33010 - 33050 |
| 33120 - 33130 |
| 33140 - 33141 |
| 33200 - 33249 |
| 33250 - 33275 |
| 33300 - 33340 |
| 33361 - 33478 |
| 33496 |
| 33500 - 33507 |
| 33600 - 33622 |
| 33641 - 33697 |
| 33702 - 33722 |
| 33724 - 33732 |
| 33735 - 33768 |
| 33770 - 33783 |
| 33786 - 33788 |
| 33800 - 33853 |
| 33860 - 33877 |
| 33880 - 33891 |
| 33910 - 33926 |
| 33962 - 33993 |
| 33999 |

| ICD-9 Procedure Codes | ICD-10 Procedure Codes |
|---|---|
| 36.91, 36.99 | 02Q00ZZ, 02Q03ZZ, 02Q04ZZ, 02Q40ZZ, 02Q43ZZ, 02Q44ZZ, 02H40YZ, 02H43YZ, 02H44YZ, 02N00ZZ, 02N03ZZ, 02N04ZZ, 02N10ZZ, 02N13ZZ, 02N14ZZ, 02N20ZZ, 02N23ZZ, 02N24ZZ, 02N30ZZ, 02N33ZZ, 02N34ZZ, 02Q00ZZ, 02Q03ZZ, 02Q04ZZ, 02Q40ZZ, 02Q43ZZ, 02Q44ZZ |
| 37.0, 37.1x, 37.3x, 37.4x, 37.5x<br>(exclude 37.51), 37.6x | 0W9D30Z, 0W9D30Z, 0W9D3ZX, 0W9D3ZX, 0W9D3ZZ, 0W9D3ZZ, 0W9D40Z, 0W9D40Z, 0W9D4ZX, 0W9D4ZX, 0W9D4ZZ, 02N60ZZ, 02N63ZZ, 02N63ZZ, 02N64ZZ, 02N6ZZZ, 02N |

| Trial ID | pNDA32 |
|---|---|
| Trial Name (with web links) | PARADIGM-HF |
| Trial Name (with pdf links) | PARADIGM-HF |
| NCT | NCT01035255 |
| Trial category | Primary indication |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | Heart failure medications |
| RCT Category | 1a- Intended S with label change |
| Brand Name | Entresto |
| Generic Name | Sacubitril/valsartan |
| <u>Sponsor</u> | Novartis |
| <u>Year</u> | 2015 |
| Measurable endpoint | Composite endpoint including death from cardiovascular causes or and hospitalization for heart failure |
| <u>Exposure</u> | LCZ696 200 mg |
| <u>Comparator</u> | Enalapril 10 mg |
| <u>Population</u> | 80% Diuretic, 29% Digitalis, 93% β blocker, 54% Mineralocorticoid antagonists, 15% ICD & 7% CRT users |
| Trial finding | HR = 0.80 (95% CI 0.73- 0.87) |
| Notes | |
| No. of Patients | 8442 |
| Non-inferiority margin | - |
| Assay Sens. Outcome | |
| Assay Sens. Endpoint (from trial) | |
| Finding for potential Assay Sens. Outcome from | |
| <u>trial-</u> | |
| <u>Power</u> | |
| Blinding | Double-blinded |
| Statistical Method | |
| Approval indication | To reduce the risk of CV death and hospitalization for heart failure in patient swith chronic heart failure (NYHA class II-IV) and reduced rejection fraction |
| אַשְאָיטימו וועונמנוטוו | reduced rejection fraction |



| | BEFORE MATCHING | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | OPTUM<br>Exposure - | | | MARKETSCAN<br>Exposure - | | | MEDICARE<br>Exposure - | | | POOLED<br>Exposure - | |
| Variable | Reference - ACE inhibitors | Sacubitril/valsartan | St. Diff | Reference - ACE inhibitors | Sacubitril/valsartan | St. Diff | Reference - ACE Inhibitors | Sacubitril/valsartan Copy | St. Diff | Reference - ACE Inhibitors | Sacubitril/valsartan Copy | St. Diff |
| Number of patients | 17,244 | 2,424 | | 10,721 | 1,289 | | 18,303 | 1,658 | | 46,268 | 5,371 | |
| Age - Continuousmean (sd) | 69.53 (11.82) | 68.49 (12.18) | 0.0867 | C2.05 (44.25) | 50.03 (43.40) | 0.2184 | 77.09 (8.22) | 76.02 (7.61) | 0.1351 | 74 22 (44 22) | 69.00 (11.33) | 0.1978 |
| mean (sd)median [IQR] | 71.00 [63.00, 78.00] | 70.00 [61.00, 78.00] | 0.0867 | 63.95 (14.26)<br>63.00 [55.00, 75.00] | 60.92 (13.48)<br>60.00 [52.00, 69.00] | 0.2184 | 76.00 [70.00, 83.00] | 75.00 [70.00, 81.00] | 0.1351 | 71.23 (11.22)<br>71.12 (11.22) | 69.14 (11.33) | 0.1978 |
| Age Categories | 71.00 [03.00, 70.00] | 70.00 [02.00, 70.00] | 0.0033 | 03.00 [33.00, 73.00] | 00.00 [32.00, 03.00] | 0.2102 | 70.00 [70.00, 03.00] | 75.00 [70.00, 01.00] | 0.1202 | 72.22 (22.22) | 03.14 (11.33) | 0.1750 |
| 18 - 54; n (%) | 1,882 (10.9%) | 332 (13.7%) | -0.0853 | 2,583 (24.1%) | 377 (29.2%) | -0.1155 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,465 (9.7%) | 709 (13.2%) | -0.1101 |
| 55 - 64; n (%)<br>65 - 74; n (%) | 3,133 (18.2%)<br>5,925 (34.4%) | 468 (19.3%)<br>807 (33.3%) | -0.0282<br>0.0232 | 3,626 (33.8%)<br>1,785 (16.6%) | 504 (39.1%)<br>169 (13.1%) | -0.1103<br>0.0985 | 0 (0.0%)<br>7,965 (43.5%) | 0 (0.0%)<br>777 (46.9%) | #DIV/0!<br>-0.0684 | 6,759 (14.6%)<br>13,890 (30.0%) | 972 (18.1%)<br>1,584 (29.5%) | -0.0947<br>0.0109 |
| 55 - 74; n (%) | 6,304 (36.6%) | 817 (33.7%) | 0.0608 | 2,727 (25.4%) | 239 (18.5%) | 0.1673 | 10,338 (56.5%) | 881 (53.1%) | 0.0684 | 16,642 (36.0%) | 1,698 (31.6%) | 0.0109 |
| Gender | | | | | | | | | | | | |
| Male; n (%) | 11,865 (68.8%) | 1,549 (63.9%) | 0.1038 | 7,721 (72.0%) | 882 (68.4%) | 0.0788 | 10,308 (56.3%) | 951 (57.4%) | -0.0222 | 22,173 (47.9%) | 2,500 (46.5%) | 0.0280 |
| Female; n (%) | 5,379 (31.2%) | 875 (36.1%) | -0.1038 | 3,000 (28.0%) | 407 (31.6%) | -0.0788 | 7,995 (43.7%) | 707 (42.6%) | 0.0222 | 13,374 (28.9%) | 1,582 (29.5%) | -0.0132 |
| Region without zero category CopyNortheast; n (%) | 2,101 (12.2%) | 273 (11.3%) | 0.0280 | 2,048 (19.1%) | 244 (18.9%) | 0.0051 | 3,372 (18.4%) | 321 (19.4%) | -0.0255 | 5,473 (11.8%) | 594 (11.1%) | 0.0220 |
| Midwest; n (%) | 8,056 (46.7%) | 1,390 (57.3%) | -0.2134 | 3,548 (33.1%) | 302 (23.4%) | 0.2167 | 7,376 (40.3%) | 771 (46.5%) | -0.1253 | 15,432 (33.4%) | 2,161 (40.2%) | -0.1414 |
| South; n (%) | 3,985 (23.1%) | 416 (17.2%) | 0.1475 | 4,096 (38.2%) | 636 (49.3%) | -0.2252 | 4,795 (26.2%) | 357 (21.5%) | 0.1105 | 8,780 (19.0%) | 773 (14.4%) | 0.1236 |
| West; n (%)Unknown+missing; n (%) | 3,086 (17.9%)<br>16 (0.1%) | 342 (14.1%)<br>3 (0.1%) | 0.1038 | 1,015 (9.5%)<br>14 (0.1%) | 106 (8.2%)<br>1 (0.1%) | 0.0458 | 2,760 (15.1%) | 209 (12.6%) | 0.0724 | 5,846 (12.6%) | 551 (10.3%) | 0.0723 |
| Calendar Time - Year of Initiation (2015/16 - 2020) | 10 (0.174) | 3 (0.1%) | 0.0000 | 14 (0.176) | 1 (0.176) | 0.0000 | | | | | | |
| 2015-2016; n (%) | 4,935 (28.6%) | 253 (10.4%) | 0.4720 | 6,045 (56.4%) | 380 (29.5%) | 0.5647 | 11,756 (64.2%) | 607 (36.6%) | 0.5743 | 16,691 (36.1%) | 860 (16.0%) | 0.4705 |
| 2017; n (%) | 3,881 (22.5%) | 500 (20.6%) | 0.0462 | 2,610 (24.3%) | 438 (34.0%) | -0.2147 | 6,547 (35.8%) | 1,051 (63.4%) | -0.5743 | 10,428 (22.5%) | 1,551 (28.9%) | -0.1469 |
| 2018; n (%)<br>2019 - 2020; n (%) | 3,960 (23.0%)<br>4,468 (25.9%) | 622 (25.7%)<br>1,049 (43.3%) | -0.0629<br>-0.3721 | 2,066 (19.3%)<br>0 (0.0%) | 471 (36.5%)<br>0 (0.0%) | -0.3907<br>#DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0!<br>#DIV/0! | 3,960 (8.6%)<br>4,468 (9.7%) | 622 (11.6%)<br>1,049 (19.5%) | -0.0997<br>-0.2802 |
| Combined comorbidity score, 180 days | 4,400 (23.5%) | 1,045 (43.376) | -0.3721 | 0 (0.0%) | 0 (0.0%) | #DIV/O: | 0 (0.0%) | 0 (0.0%) | #DIV/O: | 4,400 (3.776) | 1,043 (15.576) | -0.2802 |
| mean (sd) | 5.30 (2.55) | 5.29 (2.40) | 0.0040 | 4.21 (2.23) | 4.21 (2.12) | 0.0000 | 5.30 (2.72) | 4.75 (2.39) | 0.2148 | 5.05 (2.55) | 4.86 (2.33) | 0.0778 |
| median [IQR] | 5.00 [3.00, 7.00] | 5.00 [3.00, 7.00] | 0.0000 | 4.00 [3.00, 5.00] | 4.00 [3.00, 5.00] | 0.0000 | 5.00 [3.00, 7.00] | 4.00 [3.00, 6.00] | 0.3906 | 4.77 (2.55) | 4.45 (2.33) | 0.1310 |
| CV Comorbidity - Pulmonary hypertension/Other pulmonary heart disease ; n (%) | 2.893 (16.8%) | 506 (20.9%) | -0.1050 | 1.274 (11.9%) | 218 (16.9%) | -0.1428 | 3.611 (19.7%) | 369 (22.3%) | -0.0639 | 6.504 (14.1%) | 875 (16.3%) | -0.0613 |
| CV Comorbidity - Pulmonary hypertension/Other pulmonary heart disease; if (%) | 9,611 (55.7%) | 1,383 (57.1%) | -0.1030 | 5,648 (52.7%) | 685 (53.1%) | -0.1428 | 9,911 (54.1%) | 854 (51.5%) | 0.0521 | 19,522 (42.2%) | 2,237 (41.6%) | 0.0122 |
| CV Comorbidity - Valve disorder ; n (%) | 2,246 (13.0%) | 442 (18.2%) | -0.1437 | 657 (6.1%) | 80 (6.2%) | -0.0042 | 2,921 (16.0%) | 323 (19.5%) | -0.0917 | 5,167 (11.2%) | 765 (14.2%) | -0.0902 |
| CV Comorbidity - Hospitalization for heart failure; n (%) | 13,310 (77.2%)<br>4.746 (27.5%) | 1,891 (78.0%)<br>641 (26.4%) | -0.0192<br>0.0248 | 8,185 (76.3%)<br>2.170 (20.2%) | 971 (75.3%)<br>319 (24.7%) | 0.0234<br>-0.1080 | 15,029 (82.1%) | 1,198 (72.3%)<br>249 (15.0%) | 0.2352<br>-0.0726 | 28,339 (61.2%)<br>7.038 (15.2%) | 3,089 (57.5%) | 0.0754<br>-0.0383 |
| CV Comorbidity - Implantable cardioverter defibrillator ; n (%) CV Comorbidity - Hypotension; n (%) | 4,746 (27.5%)<br>2,300 (13.3%) | 641 (26.4%)<br>294 (12.1%) | 0.0248 | 2,170 (20.2%)<br>1,109 (10.3%) | 319 (24.7%)<br>112 (8.7%) | -0.1080<br>0.0546 | 2,292 (12.5%)<br>3,148 (17.2%) | 249 (15.0%)<br>235 (14.2%) | -0.0726<br>0.0825 | 7,038 (15.2%)<br>5,448 (11.8%) | 890 (16.6%)<br>529 (9.8%) | -0.0383<br>0.0645 |
| CV Comorbidity - Hypertension; n (%) | 15,907 (92.2%) | 2,298 (94.8%) | -0.1056 | 9,139 (85.2%) | 1,140 (88.4%) | -0.0946 | 17,177 (93.8%) | 1,591 (96.0%) | -0.1001 | 33,084 (71.5%) | 3,889 (72.4%) | -0.0200 |
| CV Comorbidity - Coronary atherosclerosis and other forms of chronic ischemic heart disease ; n (%) | 11,601 (67.3%) | 1,788 (73.8%) | -0.1430 | 6,342 (59.2%) | 753 (58.4%) | 0.0163 | 12,704 (69.4%) | 1,286 (77.6%) | -0.1866 | 24,305 (52.5%) | 3,074 (57.2%) | -0.0946 |
| CV Comorbidity - Hyperlipidemia ; n (%) CV Comorbidity - Unstable Angina (Inpatient or Outpatient) ; n (%) | 12,847 (74.5%)<br>2,054 (11.9%) | 1,968 (81.2%)<br>312 (12.9%) | -0.1619<br>-0.0303 | 6,470 (60.3%)<br>1,149 (10.7%) | 782 (60.7%)<br>126 (9.8%) | -0.0082<br>0.0297 | 13,795 (75.4%)<br>1,978 (10.8%) | 1,390 (83.8%)<br>209 (12.6%) | -0.2096<br>-0.0560 | 26,642 (57.6%)<br>4,032 (8.7%) | 3,358 (62.5%)<br>521 (9.7%) | -0.1002<br>-0.0346 |
| CV Comorbidity - Oristative Arigina (inpatient or Outpatient) ; if (%) CV Comorbidity - Implantation of CRT device: n (%) | 6.249 (36.2%) | 845 (34.9%) | 0.0272 | 3.356 (31.3%) | 457 (35.5%) | -0.0891 | 3,595 (19.6%) | 357 (21.5%) | -0.0360 | 9.844 (21.3%) | 1.202 (22.4%) | -0.0346 |
| CV Comorbidity - Stable Angina ; n (%) | 2,435 (14.1%) | 452 (18.6%) | -0.1219 | 1,114 (10.4%) | 143 (11.1%) | -0.0226 | 2,085 (11.4%) | 293 (17.7%) | -0.1794 | 4,520 (9.8%) | 745 (13.9%) | -0.1271 |
| CV Comorbidity - Stroke/TIA; n (%) | 1,680 (9.7%) | 179 (7.4%) | 0.0823 | 848 (7.9%) | 67 (5.2%) | 0.1093 | 2,531 (13.8%) | 151 (9.1%) | 0.1480 | 4,211 (9.1%) | 330 (6.1%) | 0.1134 |
| CV Comorbidity - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) CV Comorbidity - Myocardial Infarction; n (%) | 2,927 (17.0%)<br>5,921 (34.3%) | 376 (15.5%)<br>817 (33.7%) | 0.0407<br>0.0127 | 1,096 (10.2%)<br>2,982 (27.8%) | 119 (9.2%)<br>298 (23.1%) | 0.0338<br>0.1081 | 4,607 (25.2%)<br>6,043 (33.0%) | 378 (22.8%)<br>543 (32.8%) | 0.0562 | 7,534 (16.3%)<br>11,964 (25.9%) | 754 (14.0%)<br>1,360 (25.3%) | 0.0642 |
| CV Comorbidity - Myocaldan Marcton, N (%) | 8,728 (50,6%) | 1.103 (45.5%) | 0.1022 | 4.718 (44.0%) | 476 (36.9%) | 0.1450 | 10.418 (56.9%) | 870 (52.5%) | 0.0885 | 19.146 (41.4%) | 1,973 (36.7%) | 0.0965 |
| CV Comorbidity - CABG/PCI; n (%) | 5,216 (30.2%) | 865 (35.7%) | -0.1172 | 1,948 (18.2%) | 181 (14.0%) | 0.1145 | 5,049 (27.6%) | 586 (35.3%) | -0.1664 | 10,265 (22.2%) | 1,451 (27.0%) | -0.1116 |
| CONTRACTOR AND SERVICE AND | 47.244 (400.00) | 4 200 (52 40) | 1.3291 | 10,721 (100.0%) | 754 (50 704) | 1.1716 | 40 303 (400 00/) | 4.040 (54.40) | 1.1213 | 25 547 (75 00) | 2 205 (42 00) | 0.7370 |
| CV Medication - ACE inhibitors; n (%) CV Medication - Use of ARBs : n (%) | 17,244 (100.0%)<br>570 (3.3%) | 1,288 (53.1%)<br>1,271 (52.4%) | 1.3291<br>-1.3091 | 10,721 (100.0%)<br>340 (3.2%) | 764 (59.3%)<br>629 (48.8%) | -1.2169 | 18,303 (100.0%)<br>804 (4.4%) | 1,018 (61.4%)<br>727 (43.8%) | -1.0379 | 35,547 (76.8%)<br>1,374 (3,0%) | 2,306 (42.9%)<br>1.998 (37.2%) | -0.9436 |
| CV Medication - Beta blocker ; n (%) | 17,106 (99.2%) | 2,414 (99.6%) | -0.0518 | 10,629 (99.1%) | 1,284 (99.6%) | -0.0623 | 18,163 (99.2%) | 1,645 (99.2%) | 0.0000 | 35,269 (76.2%) | 4,059 (75.6%) | 0.0140 |
| CV Medication - Digoxin ; n (%) | 2,468 (14.3%) | 299 (12.3%) | 0.0589 | 1,512 (14.1%) | 187 (14.5%) | -0.0114 | 3,069 (16.8%) | 268 (16.2%) | 0.0162 | 5,537 (12.0%) | 567 (10.6%) | 0.0442 |
| CV Medication - SGLT-2 Inhibitors ; n (%) CV Medication - Loop diuretic : n (%) | 215 (1.2%)<br>13.101 (76.0%) | 82 (3.4%)<br>2.053 (84.7%) | -0.1472<br>-0.2203 | 176 (1.6%)<br>7.601 (70.9%) | 40 (3.1%)<br>1.099 (85.3%) | -0.0991<br>-0.3536 | 91 (0.5%)<br>14,036 (76,7%) | 13 (0.8%)<br>1.424 (85.9%) | -0.0373<br>-0.2376 | 306 (0.7%)<br>27.137 (58.7%) | 095 (1.8%)<br>3.477 (64.7%) | -0.0991<br>-0.1237 |
| CV Medication - Thiazide diuretics : n (%) | 13,101 (76.0%) | 2,053 (84.7%) | -0.2203 | 7,601 (70.9%)<br>957 (8.9%) | 1,099 (85.3%) | -0.3536 | 14,036 (76.7%) | 204 (12.3%) | -0.2376 | 3.074 (6.6%) | 505 (9.4%) | -0.1237 |
| CV Medication - Mineralocorticoid receptor antagonist ; n (%) | 5,642 (32.7%) | 1,112 (45.9%) | -0.2728 | 3,722 (34.7%) | 678 (52.6%) | -0.3669 | 4,839 (26.4%) | 707 (42.6%) | -0.3458 | 10,481 (22.7%) | 1,819 (33.9%) | -0.2506 |
| CV Medication - Nitrate; n (%) | 3,470 (20.1%) | 542 (22.4%) | -0.0562 | 2,113 (19.7%) | 292 (22.7%) | -0.0734 | 3,868 (21.1%) | 405 (24.4%) | -0.0788 | 7,338 (15.9%) | 947 (17.6%) | -0.0455 |
| CV Medication - PCSK9 Inhibitors; n (%) | 22 (0.1%) | 7 (0.3%) | -0.0448 | 12 (0.1%) | 5 (0.4%) | -0.0601 | 7 (0.0%) | 1 (0.1%) | -0.0447 | 029 (0.1%) | 008 (0.1%) | 0.0000 |
| CV Medication - Use of Statins ; n (%) CV Medication - Use of other lipid-lowering drugs ; n (%) | 12,062 (69.9%)<br>904 (5.2%) | 1,780 (73.4%)<br>141 (5.8%) | -0.0777<br>-0.0263 | 6,996 (65.3%)<br>600 (5.6%) | 837 (64.9%)<br>90 (7.0%) | 0.0084<br>-0.0576 | 12,124 (66.2%)<br>946 (5.2%) | 1,209 (72.9%)<br>117 (7.1%) | -0.1460<br>-0.0791 | 24,186 (52.3%)<br>1,850 (4.0%) | 2,989 (55.7%)<br>258 (4.8%) | -0.0683<br>-0.0390 |
| CV Medication - CCB (non-dihydropyridine) - Non-combo with ACEi; n (%) | 962 (5.6%) | 116 (4.8%) | 0.0360 | 573 (5.3%) | 44 (3.4%) | 0.0932 | 1,397 (7.6%) | 92 (5.5%) | 0.0850 | 2,359 (5.1%) | 208 (3.9%) | 0.0579 |
| CV Medication - CCB (dihydropyridine) - Non-combo with ACEi, ARB; n (%) | 2,589 (15.0%) | 418 (17.2%) | -0.0599 | 1,401 (13.1%) | 178 (13.8%) | -0.0205 | 3,085 (16.9%) | 263 (15.9%) | 0.0270 | 5,674 (12.3%) | 681 (12.7%) | -0.0121 |
| Other Compeliality, Otherspecies on (9) | 010 (5 200) | 125 (5 500) | 0.0400 | 202 (2.5%) | 22 /2 (2/) | 0.0000 | 1 000 (40 20) | 422 (0.00() | 0.0755 | 2 704 (5 00/) | 267 (5.004) | 0.0420 |
| Other Comorbidity - Osteoporosis ; n (%) Other Comorbidity - Dementia ; n (%) | 919 (5.3%)<br>1,767 (10.2%) | 135 (5.6%)<br>151 (6.2%) | -0.0132<br>0.1462 | 283 (2.6%)<br>672 (6.3%) | 33 (2.6%)<br>51 (4.0%) | 0.0000<br>0.1042 | 1,865 (10.2%)<br>4,311 (23.6%) | 132 (8.0%)<br>170 (10.3%) | 0.0765<br>0.3602 | 2,784 (6.0%)<br>6,078 (13.1%) | 267 (5.0%)<br>321 (6.0%) | 0.0439<br>0.2434 |
| Other Comorbidity - Dementia ; in (%) Other Comorbidity - Hypothyroidism ; n (%) | 721 (4.2%) | 87 (3.6%) | 0.0310 | 571 (5.3%) | 62 (4.8%) | 0.0228 | 1,863 (10.2%) | 97 (5.9%) | 0.1585 | 2,584 (5.6%) | 184 (3.4%) | 0.1063 |
| Other Comorbidity - Hyperthyroidism ; n (%) | 229 (1.3%) | 40 (1.7%) | -0.0329 | 148 (1.4%) | 18 (1.4%) | 0.0000 | 321 (1.8%) | 33 (2.0%) | -0.0146 | 550 (1.2%) | 073 (1.4%) | -0.0177 |
| Other Comorbidity - Hyperkalemia ; n (%) | 1,116 (6.5%)<br>2.995 (17.4%) | 150 (6.2%)<br>418 (17.2%) | 0.0123 | 445 (4.2%) | 48 (3.7%) | 0.0257 | 1,341 (7.3%)<br>4,488 (24.5%) | 97 (5.9%)<br>305 (18.4%) | 0.0564 | 2,457 (5.3%) | 247 (4.6%)<br>723 (13.5%) | 0.0323 |
| Other Comorbidity - Depression; n (%) Other Comorbidity - COPD; n (%) | 2,995 (17.4%)<br>4,922 (28.5%) | 418 (17.2%)<br>719 (29.7%) | 0.0053<br>-0.0264 | 1,184 (11.0%)<br>1,829 (17.1%) | 130 (10.1%)<br>179 (13.9%) | 0.0293 | 4,488 (24.5%)<br>5,826 (31.8%) | 305 (18.4%)<br>463 (27.9%) | 0.1490<br>0.0853 | 7,483 (16.2%)<br>10,748 (23.2%) | 723 (13.5%)<br>1,182 (22.0%) | 0.0760 |
| Other Comorbidity - Corp., IT (%) Other Comorbidity - Pneumonia; n (%) | 3,145 (18.2%) | 488 (20.1%) | -0.0483 | 1,642 (15.3%) | 215 (16.7%) | -0.0382 | 4,653 (25.4%) | 324 (19.5%) | 0.1418 | 7,798 (16.9%) | 812 (15.1%) | 0.0491 |
| Other Comorbidity - Acute kidney injury (AKI) ; n (%) | 4,102 (23.8%) | 541 (22.3%) | 0.0356 | 1,922 (17.9%) | 247 (19.2%) | -0.0334 | 5,227 (28.6%) | 375 (22.6%) | 0.1378 | 9,329 (20.2%) | 916 (17.1%) | 0.0797 |
| Other Comorbidity - CKD Stage 1-2; n (%) | 1,021 (5.9%)<br>4.224 (24.5%) | 155 (6.4%) | -0.0208<br>0.0047 | 325 (3.0%) | 29 (2.2%) | 0.0503<br>0.0211 | 1,072 (5.9%)<br>4,649 (25.4%) | 125 (7.5%) | -0.0640<br>-0.0588 | 2,093 (4.5%)<br>8,873 (19.2%) | 280 (5.2%) | -0.0326 |
| Other Comorbidity - CKD Stage 3-4; n (%) Other Comorbidity - Any Chronic Kidney Disease; n (%) | 4,224 (24.5%)<br>5,817 (33.7%) | 588 (24.3%)<br>830 (34.2%) | -0.0106 | 1,389 (13.0%)<br>1,983 (18.5%) | 159 (12.3%)<br>228 (17.7%) | 0.0211 | 4,649 (25.4%)<br>6,713 (36.7%) | 464 (28.0%)<br>639 (38.5%) | -0.0588<br>-0.0372 | 8,8/3 (19.2%)<br>12,530 (27.1%) | 1,052 (19.6%)<br>1,469 (27.4%) | -0.0101<br>-0.0067 |
| Other Comorbidity - Any Chronic Roney Disease, n (%) Other Comorbidity - Hemodialysis/Peritoneal dialysis ; n (%) | 63 (0.4%) | 6 (0.2%) | 0.0366 | 39 (0.4%) | 1 (0.1%) | 0.0601 | 88 (0.5%) | 0 (0.0%) | 0.1003 | 151 (0.3%) | 006 (0.1%) | 0.0448 |
| Other Comorbidity - DM Related Complications; n (%) | 3,822 (22.2%) | 592 (24.4%) | -0.0521 | 1,701 (15.9%) | 237 (18.4%) | -0.0664 | 4,556 (24.9%) | 409 (24.7%) | 0.0046 | 8,378 (18.1%) | 1,001 (18.6%) | -0.0129 |
| Other Comorbidity - Diabetic/Hypertensive Nephropathy; n (%) | 5,349 (31.0%) | 792 (32.7%) | -0.0365<br>-0.1232 | 1,996 (18.6%) | 266 (20.6%) | -0.0504 | 4,918 (26.9%) | 552 (33.3%) | -0.1399 | 10,267 (22.2%) | 1,344 (25.0%) | -0.0660 |
| Other Comorbidity - Sleep apnea; n (%) Other Comorbidity - Cancer : n (%) | 3,567 (20.7%)<br>2.002 (11.6%) | 628 (25.9%)<br>281 (11.6%) | 0.0000 | 2,211 (20.6%)<br>1.162 (10.8%) | 303 (23.5%)<br>108 (8.4%) | -0.0700<br>0.0815 | 2,859 (15.6%)<br>2,905 (15.9%) | 332 (20.0%)<br>228 (13.8%) | -0.1152<br>0.0591 | 6,426 (13.9%)<br>4.907 (10.6%) | 960 (17.9%)<br>509 (9.5%) | -0.1096<br>0.0366 |
| Other Comorbidity - Cancer , 11(%) Other Comorbidity - Type 1 DM ; n (%) | 648 (3.8%) | 97 (4.0%) | -0.0103 | 542 (5.1%) | 50 (3.9%) | 0.0579 | 991 (5.4%) | 72 (4.3%) | 0.0512 | 1,639 (3.5%) | 169 (3.1%) | 0.0224 |
| Other Comorbidity - Type 2 DM ; n (%) | | 1,313 (54.2%) | -0.1383 | 4,297 (40.1%) | 581 (45.1%) | -0.1012 | 8,959 (48.9%) | 852 (51.4%) | -0.0500 | 17,115 (37.0%) | 2,165 (40.3%) | -0.0678 |
| Other Comorbidity - Anemia ; n (%) | 8,156 (47.3%) | | | 2,276 (21.2%) | 250 (19.4%) | 0.0448 | 7,712 (42.1%) | 578 (34.9%) | 0.1484 | 12,324 (26.6%) | 1,241 (23.1%) | 0.0811 |
| Other Combridate Anemia , it (%) | | 663 (27.4%) | -0.0158 | -/ (/ | | | | | | | | |
| | 8,156 (47.3%) | 663 (27.4%)<br>829 (34.2%) | -0.1658 | 2.387 (22.3%) | 387 (30.0%) | -0.1759 | 3.922 (21.4%) | 399 (24.1%) | -0.0644 | 8.514 (18.4%) | 1.228 (22.9%) | -0.1113 |
| Lifestyle - Obesity ; n (%) Lifestyle - Alcohol/Drug Abuse or Dependence; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.6%) | 829 (34.2%)<br>202 (8.3%) | -0.1658<br>0.0787 | 2,387 (22.3%)<br>821 (7.7%) | 87 (6.7%) | 0.0387 | 1,365 (7.5%) | 83 (5.0%) | 0.1034 | 3,188 (6.9%) | 1,228 (22.9%)<br>285 (5.3%) | -0.1113<br>0.0669 |
| Lifestyle - Obesity ; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%) | 829 (34.2%) | -0.1658 | 2,387 (22.3%) | 387 (30.0%)<br>87 (6.7%)<br>251 (19.5%) | | | 399 (24.1%)<br>83 (5.0%)<br>681 (41.1%) | | | | |
| Lifestyle - Obesity ; n (%) Lifestyle - Alcohol/Drug Abuse or Dependence; n (%) Lifestyle - Smoking; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.6%)<br>7,970 (46.2%) | 829 (34.2%)<br>202 (8.3%)<br>1,118 (46.1%) | -0.1658<br>0.0787<br>0.0020 | 2,387 (22.3%)<br>821 (7.7%)<br>2,185 (20.4%) | 87 (6.7%)<br>251 (19.5%) | 0.0387<br>0.0225 | 1,365 (7.5%)<br>8,146 (44.5%) | 83 (5.0%)<br>681 (41.1%) | 0.1034<br>0.0688 | 3,188 (6.9%)<br>16,116 (34.8%) | 285 (5.3%)<br>1,799 (33.5%) | 0.0669<br>0.0274 |
| Lifestyle - Obesity ; n (%) Lifestyle - Alcohol/Drug Abuse or Dependence; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.6%) | 829 (34.2%)<br>202 (8.3%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149 | 2,387 (22.3%)<br>821 (7.7%)<br>2,185 (20.4%)<br>57 (0.5%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%) | 0.0387<br>0.0225<br>0.0508 | 1,365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%) | 0.1034<br>0.0688<br>0.0124 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%) | 285 (5.3%) | 0.0669<br>0.0274<br>0.0149 |
| Lifestyle - Obesity : n (%) Lifestyle - Alcoho/Drux Abuse or Dependence: n (%) Lifestyle - Snoing; n (%) Other Medication - AGI & Meglitinides ; n (%) Other Medication - Insulin; n (%) Other Medication - Cilitazones; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,512 (26.6%)<br>1,823 (10.6%)<br>7,970 (46.2%)<br>77 (0.4%)<br>2,459 (14.3%)<br>183 (1.1%) | 829 (34.2%)<br>202 (8.3%)<br>1,118 (46.1%)<br>13 (0.5%)<br>402 (16.6%)<br>34 (1.4%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149<br>-0.0637<br>-0.0270 | 2,387 (22.3%)<br>821 (7.7%)<br>2,185 (20.4%)<br>57 (0.5%)<br>1,444 (13.5%)<br>95 (0.9%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%)<br>195 (15.1%)<br>16 (1.2%) | 0.0387<br>0.0225<br>0.0508<br>-0.0457<br>-0.0294 | 1,365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%)<br>2,865 (15.7%)<br>213 (1.2%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%)<br>244 (14.7%)<br>30 (1.8%) | 0.1034<br>0.0688<br>0.0124<br>0.0279<br>-0.0494 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%)<br>5,324 (11.5%)<br>396 (0.9%) | 285 (5.3%)<br>1,799 (33.5%)<br>023 (0.4%)<br>646 (12.0%)<br>064 (1.2%) | 0.0669<br>0.0274<br>0.0149<br>-0.0155<br>-0.0294 |
| Lifestyle - Obesity : n (%) Lifestyle - Alcohol/Drug abuse or Dependence; n (%) Lifestyle - Smoking; n (%) Lifestyle - Smoking; n (%) Other Medication - AGI & Meglitinides ; n (%) Other Medication - Insulin; n (%) Other Medication - Istundranes; n (%) Other Medication - Ist and Znd Generation SUs; n (%) | 8,156 (47.3%)<br>4,512 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.5%)<br>7,970 (46.2%)<br>77 (0.4%)<br>2,459 (14.3%)<br>183 (1.1%)<br>2,076 (12.0%) | 829 (34.2%)<br>202 (8.3%)<br>1,118 (46.1%)<br>13 (0.5%)<br>402 (16.6%)<br>34 (1.4%)<br>335 (13.8%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149<br>-0.0637<br>-0.0270<br>-0.0537 | 2,387 (22.3%)<br>821 (7.7%)<br>2,185 (20.4%)<br>57 (0.5%)<br>1,444 (13.5%)<br>95 (0.9%)<br>1,133 (10.6%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%)<br>195 (15.1%)<br>16 (1.2%)<br>154 (11.9%) | 0.0387<br>0.0225<br>0.0508<br>-0.0457<br>-0.0294<br>-0.0412 | 1,365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%)<br>2,865 (15.7%)<br>213 (1.2%)<br>2,165 (11.8%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%)<br>244 (14.7%)<br>30 (1.8%)<br>242 (14.6%) | 0.1034<br>0.0688<br>0.0124<br>0.0279<br>-0.0494<br>-0.0828 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%)<br>5,324 (11.5%)<br>396 (0.9%)<br>4,241 (9.2%) | 285 (5.3%)<br>1,799 (33.5%)<br>023 (0.4%)<br>646 (12.0%)<br>064 (1.2%)<br>577 (10.7%) | 0.0669<br>0.0274<br>0.0149<br>-0.0155<br>-0.0294<br>-0.0501 |
| Lifestyle - Obesty; n (%) Lifestyle - Alcohol/Drux Abuse or Dependence: n (%) Lifestyle - Smoking; n (%) Other Medication - AGi & Meglitinides; n (%) Other Medication - Insulin; n (%) Other Medication - Cilitazones; n (%) Other Medication - Cilitazones; n (%) Other Medication - 15t and 2nd Generation SUs; n (%) Other Medication - DP-4 Inhibitors; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.6%)<br>7,970 (46.2%)<br>77 (0.4%)<br>2,459 (14.3%)<br>183 (1.1%)<br>2,076 (12.0%)<br>751 (4.4%) | 829 (34.2%) 202 (8.3%) 1,118 (46.1%) 13 (0.5%) 402 (16.6%) 34 (1.4%) 335 (13.8%) 158 (6.5%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149<br>-0.0637<br>-0.0270<br>-0.0537<br>-0.0926 | 2,387 (22,3%) 821 (7,7%) 2,185 (20,4%) 57 (0.5%) 1,444 (13.5%) 95 (0.9%) 1,133 (10.6%) 598 (5.6%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%)<br>195 (15.1%)<br>16 (1.2%)<br>154 (11.9%)<br>97 (7.5%) | 0.0387<br>0.0225<br>0.0508<br>-0.0457<br>-0.0294<br>-0.0412<br>-0.0769 | 1,365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%)<br>2,865 (15.7%)<br>213 (1.2%)<br>2,165 (11.8%)<br>935 (5.1%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%)<br>244 (14.7%)<br>30 (1.8%)<br>242 (14.6%)<br>147 (8.9%) | 0.1034<br>0.0688<br>0.0124<br>0.0279<br>-0.0494<br>-0.0828<br>-0.1493 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%)<br>5,324 (11.5%)<br>396 (0.9%)<br>4,241 (9.2%)<br>1,696 (3.7%) | 285 (5.3%)<br>1,799 (33.5%)<br>023 (0.4%)<br>646 (12.0%)<br>064 (1.2%)<br>577 (10.7%)<br>305 (5.7%) | 0.0669<br>0.0274<br>0.0149<br>-0.0155<br>-0.0294<br>-0.0501<br>-0.0946 |
| Lifestyle - Obestty : n (%) Lifestyle - Alcohol/Orus Abuse or Dependence; n (%) Lifestyle - Smoking; n (%) Lifestyle - Smoking; n (%) Other Medication - AGI & Meglitinides ; n (%) Other Medication - Insulin; n (%) Other Medication - Insulin; n (%) Other Medication - Ist and Znd Generation SUs; n (%) Other Medication - 184 and Znd Generation SUs; n (%) Other Medication - 184 and Znd Generation SUs; n (%) Other Medication - GEP-18 n; n (%) | 8.156 (47.3%)<br>4,612 (26.7%)<br>4,512 (26.6%)<br>1,823 (10.6%)<br>7,970 (46.2%)<br>77 (0.4%)<br>2,459 (14.3%)<br>183 (1.1%)<br>2,076 (12.0%)<br>761 (4.4%)<br>326 (1.9%) | 829 (34.2%) 202 (8.3%) 1,118 (46.1%) 13 (0.5%) 402 (16.6%) 34 (1.4%) 335 (13.8%) 158 (6.5%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149<br>-0.0637<br>-0.0270<br>-0.0537<br>-0.0926<br>-0.1341 | 2,387 (22.3%) 821 (7.7%) 2,185 (20.4%) 57 (0.5%) 1,444 (13.5%) 95 (0.9%) 1,133 (10.6%) 598 (5.6%) 210 (2.0%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%)<br>195 (15.1%)<br>16 (1.2%)<br>154 (11.9%)<br>97 (7.5%)<br>47 (3.6%) | 0.0387<br>0.0225<br>0.0508<br>-0.0457<br>-0.0294<br>-0.0412<br>-0.0769<br>-0.0971 | 1,365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%)<br>2,865 (15.7%)<br>213 (1.2%)<br>2,165 (11.8%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%)<br>244 (14.7%)<br>30 (1.8%)<br>242 (14.6%)<br>147 (8.9%)<br>24 (1.4%) | 0.1034<br>0.0688<br>0.0124<br>0.0279<br>-0.0494<br>-0.0828 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%)<br>5,324 (11.5%)<br>396 (0.9%)<br>4,241 (9.2%)<br>1,696 (3.7%)<br>477 (1.0%) | 285 (5.3%)<br>1,799 (33.5%)<br>023 (0.4%)<br>646 (12.0%)<br>064 (1.2%)<br>577 (10.7%)<br>305 (5.7%)<br>125 (2.3%) | 0.0669<br>0.0274<br>0.0149<br>-0.0155<br>-0.0294<br>-0.0501<br>-0.0946<br>-0.1022 |
| Lifestyle - Obesty; n (%) Lifestyle - Alcohol/Drux Abuse or Dependence: n (%) Lifestyle - Smoking; n (%) Other Medication - AGi & Meglitinides; n (%) Other Medication - Insulin; n (%) Other Medication - Cilitazones; n (%) Other Medication - Cilitazones; n (%) Other Medication - 15t and 2nd Generation SUs; n (%) Other Medication - DP-4 Inhibitors; n (%) | 8,156 (47.3%)<br>4,612 (26.7%)<br>4,592 (26.6%)<br>1,823 (10.6%)<br>7,970 (46.2%)<br>77 (0.4%)<br>2,459 (14.3%)<br>183 (1.1%)<br>2,076 (12.0%)<br>751 (4.4%) | 829 (34.2%) 202 (8.3%) 1,118 (46.1%) 13 (0.5%) 402 (16.6%) 34 (1.4%) 335 (13.8%) 158 (6.5%) | -0.1658<br>0.0787<br>0.0020<br>-0.0149<br>-0.0637<br>-0.0270<br>-0.0537<br>-0.0926 | 2,387 (22,3%) 821 (7,7%) 2,185 (20,4%) 57 (0.5%) 1,444 (13.5%) 95 (0.9%) 1,133 (10.6%) 598 (5.6%) | 87 (6.7%)<br>251 (19.5%)<br>3 (0.2%)<br>195 (15.1%)<br>16 (1.2%)<br>154 (11.9%)<br>97 (7.5%) | 0.0387<br>0.0225<br>0.0508<br>-0.0457<br>-0.0294<br>-0.0412<br>-0.0769 | 1.365 (7.5%)<br>8,146 (44.5%)<br>132 (0.7%)<br>2,865 (15.7%)<br>213 (1.2%)<br>2,165 (11.8%)<br>935 (5.1%)<br>151 (0.8%) | 83 (5.0%)<br>681 (41.1%)<br>10 (0.6%)<br>244 (14.7%)<br>30 (1.8%)<br>242 (14.6%)<br>147 (8.9%) | 0.1034<br>0.0688<br>0.0124<br>0.0279<br>-0.0494<br>-0.0828<br>-0.1493<br>-0.0575 | 3,188 (6.9%)<br>16,116 (34.8%)<br>209 (0.5%)<br>5,324 (11.5%)<br>396 (0.9%)<br>4,241 (9.2%)<br>1,696 (3.7%) | 285 (5.3%)<br>1,799 (33.5%)<br>023 (0.4%)<br>646 (12.0%)<br>064 (1.2%)<br>577 (10.7%)<br>305 (5.7%) | 0.0669<br>0.0274<br>0.0149<br>-0.0155<br>-0.0294<br>-0.0501<br>-0.0946 |

| Other Medication - Use of antiplatelet agents ; n (%) | 4.412 (25.6%) | 695 (28.7%) | -0.0697 | 3.239 (30.2%) | 404 (31.3%) | -0.0238 | 4.061 (22.2%) | 466 (28.1%) | -0.1363 | 8.473 (18.3%) | 1.161 (21.6%) | -0.0826 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Other Medication - Use of Antiplateiet agents , if (%) Other Medication - Use of heparin and other low-molecular weight heparins ; n (%) | 370 (2.1%) | 42 (1.7%) | 0.0293 | 6 (0.1%) | 0 (0.0%) | 0.0447 | 472 (2.6%) | 18 (1.1%) | 0.1115 | 842 (1.8%) | 060 (1.1%) | 0.0586 |
| Other Medication - Use of oral anticoagulants ; n (%) | 6,844 (39.7%) | 935 (38.6%) | 0.0225 | 4,175 (38.9%) | 471 (36.5%) | 0.0495 | 7,403 (40.4%) | 690 (41.6%) | -0.0244 | 14,247 (30.8%) | 1,625 (30.3%) | 0.0109 |
| Other Medication - Use of other hypertension drugs; n (%) | 1,923 (11.2%) | 300 (12.4%) | -0.0372 | 1,199 (11.2%) | 179 (13.9%) | -0.0816 | 2,063 (11.3%) | 202 (12.2%) | -0.0280 | 3,986 (8.6%) | 502 (9.3%) | -0.0245 |
| Other Medication - Use of antipsychotics ; n (%) | 541 (3.1%) | 60 (2.5%) | 0.0364 | 233 (2.2%) | 22 (1.7%) | 0.0362 | 1.073 (5.9%) | 46 (2.8%) | 0.1524 | 1.614 (3.5%) | 106 (2.0%) | 0.0918 |
| Other Medication - Use of dementia meds : n (%) | 518 (3.0%) | 50 (2.1%) | 0.0571 | 216 (2.0%) | 21 (1.6%) | 0.0301 | 1,295 (7.1%) | 66 (4.0%) | 0.1357 | 1.813 (3.9%) | 116 (2.2%) | 0.0990 |
| Other Medication - Use of antiparkinsonian meds : n (%) | 435 (2.5%) | 74 (3.1%) | -0.0364 | 189 (1.8%) | 28 (2.2%) | -0.0286 | 741 (4.0%) | 45 (2.7%) | 0.0723 | 1.176 (2.5%) | 119 (2.2%) | 0.0198 |
| Other Medication - Use of anxiolytics/hypnotics; n (%) | 1,014 (5.9%) | 159 (6.6%) | -0.0289 | 671 (6.3%) | 85 (6.6%) | -0.0122 | 1,137 (6.2%) | 123 (7.4%) | -0.0477 | 2,151 (4.6%) | 282 (5.3%) | -0.0323 |
| Other Medication - Use of anticonvulsants ; n (%) | 3,043 (17.6%) | 403 (16.6%) | 0.0266 | 1,319 (12.3%) | 137 (10.6%) | 0.0534 | 3,713 (20.3%) | 267 (16.1%) | 0.1090 | 6,756 (14.6%) | 670 (12.5%) | 0.0614 |
| Other Medication - Use of antidepressants ; n (%) | 4,418 (25.6%) | 618 (25.5%) | 0.0023 | 2,297 (21.4%) | 266 (20.6%) | 0.0196 | 5,702 (31.2%) | 454 (27.4%) | 0.0836 | 10,120 (21.9%) | 1,072 (20.0%) | 0.0467 |
| Other Medication - Use of lithium ; n (%) | 14 (0.1%) | 2 (0.1%) | 0.0000 | 16 (0.1%) | 0 (0.0%) | 0.0447 | 16 (0.1%) | 0 (0.0%) | 0.0447 | 030 (0.1%) | 002 (0.0%) | 0.0447 |
| Other Medication - Use of Benzodiazepine; n (%) | 2,208 (12.8%) | 328 (13.5%) | -0.0207 | 1,321 (12.3%) | 184 (14.3%) | -0.0589 | 2,763 (15.1%) | 257 (15.5%) | -0.0111 | 4,971 (10.7%) | 585 (10.9%) | -0.0064 |
| Other Medication - Use of opioids ; n (%) | 5,405 (31.3%) | 712 (29.4%) | 0.0413 | 3,310 (30.9%) | 336 (26.1%) | 0.1065 | 6,255 (34.2%) | 447 (27.0%) | 0.1567 | 11,660 (25.2%) | 1,159 (21.6%) | 0.0851 |
| Other Medication - Use of COPD/asthma meds ; n (%) | 3,139 (18.2%) | 549 (22.6%) | -0.1094 | 1,703 (15.9%) | 265 (20.6%) | -0.1219 | 3,142 (17.2%) | 358 (21.6%) | -0.1114 | 6,281 (13.6%) | 907 (16.9%) | -0.0919 |
| HU - Bone mineral density; n (%) | 348 (2.0%) | 56 (2.3%) | -0.0207 | 99 (0.9%) | 17 (1.3%) | -0.0384 | 364 (2.0%) | 31 (1.9%) | 0.0072 | 712 (1.5%) | 087 (1.6%) | -0.0081 |
| HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) | 646 (3.7%) | 86 (3.5%) | 0.0107 | 440 (4.1%) | 54 (4.2%) | -0.0050 | 789 (4.3%) | 63 (3.8%) | 0.0254 | 1,435 (3.1%) | 149 (2.8%) | 0.0177 |
| HU - Flu vaccine; n (%) | 2,851 (16.5%) | 446 (18.4%) | -0.0501 | 1,106 (10.3%) | 142 (11.0%) | -0.0227 | 4,410 (24.1%) | 491 (29.6%) | -0.1243 | 7,261 (15.7%) | 937 (17.4%) | -0.0458 |
| HU - Mammogram; n (%) | 775 (4.5%) | 135 (5.6%) | -0.0503 | 404 (3.8%) | 62 (4.8%) | -0.0493 | 830 (4.5%) | 88 (5.3%) | -0.0371 | 1,605 (3.5%) | 223 (4.2%) | -0.0364 |
| HU - Frailty Score: Empirical Version 365 days | | | | | | | | | | | | |
| mean (sd) | 0.23 (0.07) | 0.22 (0.06) | 0.1534 | 0.20 (0.06) | 0.20 (0.05) | 0.0000 | 0.27 (0.09) | 0.24 (0.07) | 0.3721 | 0.24 (0.08) | 0.22 (0.06) | 0.2828 |
| median [IQR] | 0.21 [0.18, 0.26] | 0.21 [0.18, 0.25] | 0.0000 | 0.19 [0.16, 0.23] | 0.19 [0.16, 0.21] | 0.0000 | 0.25 [0.20, 0.32] | 0.23 [0.19, 0.27] | 0.2481 | 0.22 (0.08) | 0.21 (0.06) | 0.1414 |
| HU - Number of hospitalizations during CAP | | | | | | | | | | | | |
| mean (sd) | 1.06 (0.84) | 1.03 (0.76) | 0.0375 | 0.96 (0.74) | 0.90 (0.68) | 0.0844 | 1.39 (1.10) | 1.04 (0.89) | 0.3498 | 1.17 (0.93) | 1.00 (0.78) | 0.1981 |
| median [IQR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 2.00] | 1.00 [0.00, 1.00] | 0.0000 | 1.00 (0.93) | 1.00 (0.78) | 0.0000 |
| HU - Number of Emergency Department (ED) visits | | | | | | | | | | | | |
| mean (sd) | 1.71 (2.73) | 1.79 (2.36) | -0.0314 | 2.23 (4.68) | 2.17 (3.64) | 0.0143 | 2.07 (2.66) | 1.59 (2.55) | 0.1842 | 1.97 (3.26) | 1.82 (2.77) | 0.0496 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.00 [0.00, 3.00] | 0.00 [0.00, 3.00] | 0.0000 | 1.00 [0.00, 3.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.77 (3.26) | 0.76 (2.77) | 0.0033 |
| HU - Number of Internal Medicine/Family Medicine Visits | | | | | | | | | | | | |
| mean (sd) | 14.57 (17.87)<br>9.00 [4.00, 19.00] | 14.29 (17.89)<br>9.00 [4.00, 19.00] | 0.0157 | 9.73 (14.69)<br>5.00 [2.00, 12.00] | 9.03 (13.38)<br>5.00 [2.00, 11.00] | 0.0498 | 12.75 (15.11) | 8.88 (11.78)<br>6.00 [3.00, 11.00] | 0.2857<br>0.1476 | 12.73 (16.10)<br>7.68 (16.10) | 11.36 (15.17) | 0.0876 |
| median [IQR] HU - Number of Distinct Medication Prescriptions (not generalized to generics) | 9.00 [4.00, 19.00] | 9.00 [4.00, 19.00] | 0.0000 | 5.00 [2.00, 12.00] | 5.00 [2.00, 11.00] | 0.0000 | 8.00 [4.00, 16.00] | 6.00 [3.00, 11.00] | 0.1476 | 7.68 (16.10) | 7.11 (15.17) | 0.0364 |
| mean (sd) | 30.67 (20.95) | 34.27 (21.45) | -0.1698 | 25.34 (13.88) | 30.86 (15.63) | -0.3735 | 27.59 (17.12) | 33.01 (17.68) | -0.3115 | 28.22 (18.00) | 33.06 (19.05) | -0.2612 |
| median (IQR) | 26.00 [17.00, 38.00] | 30.00 [20.00, 42.00] | -0.1887 | 23.00 [16.00, 32.00] | 28.00 [20.00, 38.00] | -0.3383 | 24.00 [16.00, 35.00] | 29.00 [21.00, 40.00] | -0.2873 | 24.51 (18.00) | 29.21 (19.05) | -0.2536 |
| median [iQK] HU - Number of Cardiologist visits | 26.00 [17.00, 38.00] | 30.00 [20.00, 42.00] | -0.1887 | 23.00 [16.00, 32.00] | 28.00 [20.00, 38.00] | -0.3383 | 24.00 [16.00, 35.00] | 29.00 [21.00, 40.00] | -0.28/3 | 24.51 (18.00) | 29.21 (19.05) | -0.2536 |
| mean (sd) | 10.80 (10.03) | 13.40 (10.60) | -0.2520 | 5.27 (7.42) | 7.15 (7.98) | -0.2440 | 8.94 (9.61) | 11.44 (11.32) | -0.2381 | 8.78 (9.32) | 11.30 (10.27) | -0.2570 |
| median [IQR] | 8.00 [4.00, 15.00] | 11.00 [6.00, 18.00] | -0.2907 | 3.00 [0.00, 8.00] | 5.00 [2.00, 10.00] | -0.2596 | 6.00 [2.00, 12.00] | 9.00 [4.00, 15.00] | -0.2351 | 6.05 (9.32) | 8.94 (10.27) | -0.2947 |
| HU - Number of Electrocardiogram | 5.00 [4.00, 15.00] | 11.00 [0.00, 10.00] | 0.2307 | 5.50 [5.50, 8.50] | 3.55 [2.50, 10.50] | 0.2390 | 0.00 [2.00, 12.00] | 3.00 [4.00, 13.00] | 0.2037 | 0.03 (3.32) | 0.54 (10.27) | 0.2347 |
| mean (sd) | 3.68 (3.91) | 4.18 (4.12) | -0.1245 | 2.90 (2.79) | 3.12 (2.87) | -0.0777 | 3.42 (3.25) | 3.63 (3.59) | -0.0613 | 3.40 (3.42) | 3.76 (3.69) | -0.1012 |
| median [JQR] | 3.00 (1.00, 5.00) | 3.00 [2.00, 6.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 3.00 [1.00, 5.00] | 3.00 [1.00, 5.00] | 0.0000 | 2.77 (3.42) | 2.76 (3.69) | 0.0028 |
| HU - Number of Echocardiogram | 3.00 [2.00, 3.00] | 5.00 [2.00, 0.00] | 0.0000 | 00 [2.00, 4.00] | 2.00 [2.00, 7.00] | 0.0000 | 3.00 [2.00, 3.00] | 3.00 [2.00, 3.00] | 0.0000 | 2.77 (3.72) | 2.70 (3.03) | 0.0020 |
| mean (sd) | 2.28 (5.02) | 2.58 (4.76) | -0.0613 | 1.52 (1.70) | 1.66 (1.59) | -0.0851 | 1.33 (1.25) | 1.60 (1.40) | -0.2034 | 1.73 (3.27) | 2.06 (3.38) | -0.0992 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [1.00, 3.00] | 0.0000 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.0000 | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.0000 | 1.00 (3.27) | 1.00 (3.38) | 0.0000 |
| SES Proxy - Copay for pharmacy cost (charges in U.S. \$) | ( , , | | | , , , , , , | ,,, | 1 | | ,, | | ,, | . (0.00) | |
| mean (sd) | 24.10 (34.04) | 26.12 (30.50) | -0.0625 | 14.67 (18.89) | 15.10 (17.86) | -0.0234 | 22.05 (33.42) | 26.07 (29.82) | -0.1269 | 21.10 (30.93) | 23.46 (27.77) | -0.0803 |
| median [IQR] | 14.62 [5.79, 30.27] | 18.66 [6.73, 34.59] | -0.1250 | 10.46 [3.57, 19.54] | 12.42 [4.76, 20.28] | -0.1066 | 12.90 [4.04, 28.02] | 18.49 [5.40, 34.97] | -0.1765 | 12.98 (30.93) | 17.11 (27.77) | -0.1405 |
| SES Proxy - Low income indicator: n (%) | 3,942 (22.9%) | 541 (22.3%) | 0.0143 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3.942 (8.5%) | 541 (10.1%) | -0.0551 |
| SES Proxy - Business type | .,. (===,-, | , (-2.07.7) | ,,,,,,, | . 1 | . (5.5.5) | 11,701 | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | . ( | .,,, | .,. (0.012) | . ( | |
| Commercial: n (%) | 3,171 (18.4%) | 610 (25.2%) | -0.1653 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3.171 (6.9%) | 610 (11.4%) | -0.1566 |
| Medicare: n (%) | 14.073 (81.6%) | 1.814 (74.8%) | 0.1653 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 14.073 (30.4%) | 1.814 (33.8%) | -0.0729 |
| SES Proxy - Insurance Plan type | ,(04.07.7) | ,. (************************************ | | . 1 | . (5.5.5) | , | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | . ( | .,,, | ,, | , (44,4,4) | |
| Comprehensive; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,527 (23.6%) | 175 (13.6%) | 0.2591 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,527 (5.5%) | 175 (3.3%) | 0.1074 |
| HMO; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,060 (9.9%) | 112 (8.7%) | 0.0413 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 1,060 (2.3%) | 112 (2.1%) | 0.0136 |
| PPO; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,951 (46.2%) | 686 (53.2%) | -0.1403 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,951 (10.7%) | 686 (12.8%) | -0.0652 |
| Others; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,183 (20.4%) | 316 (24.5%) | -0.0984 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 2,183 (4.7%) | 316 (5.9%) | -0.0536 |
| SES Proxy - Dual status code (with Medicaid); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 4,785 (26.1%) | 343 (20.7%) | 0.1278 | 4,785 (10.3%) | 343 (6.4%) | 0.1413 |
| | . , | . ,,,,,,,,,, | , | . () | . (0.0) | ,, | , (2002) | , , | | , (-0.0.1) | , | |

| | AFTER MATCHING OPTUM MARKETSCAN MEDICARE POOLED | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Reference - ACE | | Reference - ACE | MARKETSCAN Exposure - | | Reference - ACE | MEDICARE<br>Exposure - | | Reference - ACE | POOLED<br>Exposure - | | |
| | inhibitors | Exposure -<br>Sacubitril/valsartan | St. Diff | inhibitors | Sacubitril/valsartan | St. Diff | Inhibitors | Sacubitril/valsartan | St. Diff | Inhibitors | Sacubitril/valsartan | St. Diff |
| Number of patients | 1,279 | 1,279 | | 748 | 748 | | 1,006 | 1,006 | I | 3,033 | 3,033 | |
| Age - Continuousmean (sd) | 68.68 (11.85) | 67.91 (12.31) | 0.0637 | 59.59 (13.80) | 60.00 (13.63) | -0.0299 | 75.41 (7.47) | 75.61 (7.51) | -0.0267 | 68.67 (11.17) | 68.51 (11.33) | 0.0142 |
| median [IQR] | 69.00 [61.00, 77.00] | 69.00 [60.00, 77.00] | 0.0000 | 58.50 [51.00, 68.00] | 60.00 [52.00, 68.00] | -0.1094 | 74.00 [69.00, 81.00] | 75.00 [69.00, 81.00] | -0.1335 | 68.07 (11.17) | 68.77 (11.33) | -0.0622 |
| Age Categories* | 137 (10.7%) | 196 (15.3%) | -0.1371 | 262 (25 20/) | 236 (31.6%) | 0.0764 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 400 (13.2%) | 432 (14.2%) | -0.0291 |
| 18 - 54; n (%)<br>55 - 64; n (%) | 285 (22.3%) | 256 (20.0%) | 0.0563 | 263 (35.2%)<br>265 (35.4%) | 284 (38.0%) | -0.0540 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 550 (18.1%) | 540 (17.8%) | 0.0078 |
| 65 - 74; n (%) | 427 (33.4%) | 411 (32.1%) | 0.0277 | 111 (14.8%) | 103 (13.8%) | 0.0286 | 514 (51.1%) | 492 (48.9%) | 0.0440 | 941 (31.0%) | 903 (29.8%) | 0.0261 |
| >= 75; n (%) | 430 (33.6%) | 416 (32.5%) | 0.0234 | 109 (14.6%) | 125 (16.7%) | -0.0578 | 492 (48.9%) | 514 (51.1%) | -0.0440 | | | |
| GenderMale: n (%) | 880 (68.8%) | 855 (66.8%) | 0.0428 | 541 (72.3%) | 535 (71.5%) | 0.0178 | 589 (58.5%) | 604 (60.0%) | -0.0305 | 1,469 (48.4%) | 1,459 (48.1%) | 0.0060 |
| Female; n (%) | 399 (31.2%) | 424 (33.2%) | -0.0428 | 207 (27.7%) | 213 (28.5%) | -0.0178 | 417 (41.5%) | 402 (40.0%) | 0.0305 | 816 (26.9%) | 826 (27.2%) | -0.0068 |
| Region without zero categoryNortheast; n (%) | 142 (11.1%) | 140 (10.9%) | 0.0064 | 137 (18.3%) | 142 (19.0%) | -0.0180 | 159 (15.8%) | 195 (19.4%) | -0.0946 | 301 (9.9%) | 335 (11.0%) | -0.0360 |
| Notuteast, it (%) | 722 (56.5%) | 715 (55.9%) | 0.0004 | 202 (27.0%) | 180 (24.1%) | 0.0665 | 482 (47.9%) | 469 (46.6%) | 0.0260 | 1,204 (39.7%) | 1,184 (39.0%) | 0.0143 |
| South; n (%) | 227 (17.7%) | 247 (19.3%) | -0.0412 | 370 (49.5%) | 366 (48.9%) | 0.0120 | 232 (23.1%) | 221 (22.0%) | 0.0263 | 459 (15.1%) | 468 (15.4%) | -0.0083 |
| West; n (%)Unknown+missing; n (%) | 188 (14.7%) | 177 (13.8%)<br>0 (0.0%) | 0.0257<br>#DIV/0! | 39 (5.2%)<br>0 (0.0%) | 60 (8.0%)<br>0 (0.0%) | -0.1130<br>#DIV/0! | 133 (13.2%) | 121 (12.0%) | 0.0362 | 321 (10.6%) | 298 (9.8%) | 0.0264 |
| Calendar Time - Year of Initiation (2015/16 - 2020) | 0 (0.0%) | 0 (0.0%) | #DIV/U: | 0 (0.0%) | 0 (0.0%) | #010/0: | | | + | | | + |
| 2015-2016; n (%) | 146 (11.4%) | 153 (12.0%) | -0.0187 | 229 (30.6%) | 233 (31.1%) | -0.0108 | 355 (35.3%) | 374 (37.2%) | -0.0395 | 797 (26.3%) | 785 (25.9%) | 0.0091 |
| 2017; n (%)<br>2018; n (%) | 293 (22.9%)<br>321 (25.1%) | 280 (21.9%)<br>319 (24.9%) | 0.0240<br>0.0046 | 264 (35.3%)<br>255 (34.1%) | 256 (34.2%)<br>259 (34.6%) | 0.0231<br>-0.0105 | 651 (64.7%)<br>0 (0.0%) | 632 (62.8%)<br>0 (0.0%) | 0.0395<br>#DIV/0! | 293 (9.7%)<br>321 (10.6%) | 280 (9.2%)<br>319 (10.5%) | 0.0171<br>0.0033 |
| 2019 - 2020; n (%) | 519 (40.6%) | 527 (41.2%) | -0.0122 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 519 (40.6%) | 527 (41.2%) | -0.0122 |
| Combined comorbidity score, 180 days | | | | .,, | | | | .,, | | | | |
| mean (sd)median [IQR] | 5.30 (2.47)<br>5.00 [4.00, 7.00] | 5.27 (2.43)<br>5.00 [3.00, 7.00] | 0.0122 | 4.24 (2.12)<br>4.00 [3.00, 6.00] | 4.19 (2.06)<br>4.00 [3.00, 5.00] | 0.0239 | 4.77 (2.49)<br>4.00 [3.00, 6.00] | 4.76 (2.40)<br>4.00 [3.00, 6.00] | 0.0041 | 4.86 (2.40)<br>4.42 (2.40) | 4.83 (2.33)<br>4.42 (2.33) | 0.0127 |
| amedian papa | | | 0.0000 | 00 [5.00, 0.00] | 4.00 [3.00, 3.00] | 0.000 | 00 [5.00, 0.00] | 00 [5.00, 0.00] | | 4.42 (2.40) | 4.42 (2.33) | 3.000 |
| CV Comorbidity - Pulmonary hypertension/Other pulmonary heart disease ; n (%) | 250 (19.5%) | 257 (20.1%) | -0.0151 | 132 (17.6%) | 126 (16.8%) | 0.0212 | 209 (20.8%) | 223 (22.2%) | -0.0341 | 459 (15.1%) | 480 (15.8%) | -0.0194 |
| CV Comorbidity - Other dysrythmias ; n (%) | 735 (57.5%)<br>254 (19.9%) | 736 (57.5%)<br>237 (18.5%) | 0.0000 | 424 (56.7%)<br>46 (6.1%) | 409 (54.7%)<br>49 (6.6%) | 0.0403<br>-0.0205 | 506 (50.3%)<br>202 (20.1%) | 519 (51.6%)<br>203 (20.2%) | -0.0260<br>-0.0025 | 1,241 (40.9%)<br>456 (15.0%) | 1,255 (41.4%)<br>440 (14.5%) | -0.0102<br>0.0141 |
| CV Comorbidity - Valve disorder ; n (%) CV Comorbidity - Hospitalization for heart failure; n (%) | 1,041 (81.4%) | 1,051 (82.2%) | -0.0207 | 602 (80.5%) | 593 (79.3%) | 0.0299 | 743 (73.9%) | 740 (73.6%) | 0.0068 | 1,784 (58.8%) | 1,791 (59.1%) | -0.0061 |
| CV Comorbidity - Implantable cardioverter defibrillator ; n (%) | 328 (25.6%) | 303 (23.7%) | 0.0441 | 170 (22.7%) | 170 (22.7%) | 0.0000 | 137 (13.6%) | 145 (14.4%) | -0.0231 | 465 (15.3%) | 448 (14.8%) | 0.0140 |
| CV Comorbidity - Hypotension; n (%) CV Comorbidity - Hypertension; n (%) | 167 (13.1%)<br>1,206 (94.3%) | 169 (13.2%)<br>1,208 (94.4%) | -0.0030<br>-0.0043 | 67 (9.0%)<br>666 (89.0%) | 73 (9.8%)<br>658 (88.0%) | -0.0274<br>0.0313 | 160 (15.9%)<br>972 (96.6%) | 150 (14.9%)<br>960 (95.4%) | 0.0277<br>0.0613 | 327 (10.8%)<br>2,178 (71.8%) | 319 (10.5%)<br>2,168 (71.5%) | 0.0097<br>0.0067 |
| CV Comorbidity - Tryperterision, it (%) CV Comorbidity - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 959 (75.0%) | 946 (74.0%) | 0.0229 | 436 (58.3%) | 427 (57.1%) | 0.0243 | 780 (77.5%) | 788 (78.3%) | -0.0193 | 1,739 (57.3%) | 1,734 (57.2%) | 0.0020 |
| CV Comorbidity - Hyperlipidemia ; n (%) | 1,026 (80.2%) | 1,020 (79.7%) | 0.0125 | 446 (59.6%) | 446 (59.6%) | 0.0000 | 830 (82.5%) | 835 (83.0%) | -0.0132 | 1,856 (61.2%) | 1,855 (61.2%) | 0.0000 |
| CV Comorbidity - Unstable Angina (Inpatient or Outpatient) ; n (%) CV Comorbidity - Implantation of CRT device; n (%) | 161 (12.6%)<br>428 (33.5%) | 173 (13.5%)<br>409 (32.0%) | -0.0267<br>0.0320 | 78 (10.4%)<br>239 (32.0%) | 81 (10.8%)<br>239 (32.0%) | -0.0130<br>0.0000 | 146 (14.5%)<br>193 (19.2%) | 139 (13.8%)<br>205 (20.4%) | 0.0201<br>-0.0301 | 307 (10.1%)<br>621 (20.5%) | 312 (10.3%)<br>614 (20.2%) | -0.0066<br>0.0075 |
| CV Comorbidity - Stable Angina ; n (%) | 232 (18.1%) | 241 (18.8%) | -0.0180 | 94 (12.6%) | 79 (10.6%) | 0.0625 | 203 (20.2%) | 184 (18.3%) | 0.0482 | 435 (14.3%) | 425 (14.0%) | 0.0086 |
| CV Comorbidity - Stroke/TIA; n (%) | 81 (6.3%) | 101 (7.9%) | -0.0623 | 44 (5.9%) | 45 (6.0%) | -0.0042 | 83 (8.3%) | 90 (8.9%) | -0.0214 | 164 (5.4%) | 191 (6.3%) | -0.0384 |
| CV Comorbidity - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) CV Comorbidity - Myocardial Infarction; n (%) | 192 (15.0%)<br>450 (35.2%) | 189 (14.8%)<br>447 (34.9%) | 0.0056<br>0.0063 | 69 (9.2%)<br>190 (25.4%) | 68 (9.1%)<br>182 (24.3%) | 0.0035<br>0.0255 | 230 (22.9%)<br>363 (36.1%) | 238 (23.7%)<br>362 (36.0%) | -0.0189<br>0.0021 | 422 (13.9%)<br>813 (26.8%) | 427 (14.1%)<br>809 (26.7%) | -0.0058<br>0.0023 |
| CV Comorbidity - Atrial fibrillation; n (%) | 576 (45.0%) | 562 (43.9%) | 0.0221 | 258 (34.5%) | 275 (36.8%) | -0.0480 | 537 (53.4%) | 524 (52.1%) | 0.0260 | 1,113 (36.7%) | 1,086 (35.8%) | 0.0187 |
| CV Comorbidity - CABG/PCI; n (%) | 478 (37.4%) | 478 (37.4%) | 0.0000 | 142 (19.0%) | 120 (16.0%) | 0.0790 | 369 (36.7%) | 374 (37.2%) | -0.0104 | 847 (27.9%) | 852 (28.1%) | -0.0045 |
| CV Medication - ACE inhibitors: n (%) | 1.279 (100.0%) | 1.279 (100.0%) | #DIV/0! | 748 (100.0%) | 748 (100.0%) | #DIV/0! | 1.006 (100.0%) | 1.006 (100.0%) | #DIV/0! | 2.285 (75.3%) | 2.285 (75.3%) | 0.0000 |
| CV Medication - Use of ARBs ; n (%) | 118 (9.2%) | 127 (9.9%) | -0.0238 | 92 (12.3%) | 89 (11.9%) | 0.0123 | 75 (7.5%) | 81 (8.1%) | -0.0224 | 193 (6.4%) | 208 (6.9%) | -0.0201 |
| CV Medication - Beta blocker ; n (%) | 1,273 (99.5%)<br>162 (12.7%) | 1,273 (99.5%)<br>158 (12.4%) | 0.0000 | 747 (99.9%)<br>104 (13.9%) | 746 (99.7%)<br>106 (14.2%) | 0.0448<br>-0.0086 | 998 (99.2%)<br>172 (17.1%) | 999 (99.3%)<br>160 (15.9%) | -0.0116<br>0.0323 | 2,271 (74.9%)<br>334 (11.0%) | 2,272 (74.9%)<br>318 (10.5%) | 0.0000<br>0.0161 |
| CV Medication - Digoxin ; n (%) CV Medication - SGLT-2 Inhibitors ; n (%) | 48 (3.8%) | 42 (3.3%) | 0.0091 | 18 (2.4%) | 22 (2.9%) | -0.0086 | 2 (0.2%) | 5 (0.5%) | -0.0508 | 050 (1.6%) | 047 (1.5%) | 0.0161 |
| CV Medication - Loop diuretic ; n (%) | 1,078 (84.3%) | 1,081 (84.5%) | -0.0055 | 645 (86.2%) | 637 (85.2%) | 0.0286 | 880 (87.5%) | 859 (85.4%) | 0.0614 | 1,958 (64.6%) | 1,940 (64.0%) | 0.0125 |
| CV Medication - Thiazide diuretics ; n (%) | 147 (11.5%) | 155 (12.1%) | -0.0186 | 82 (11.0%) | 88 (11.8%) | -0.0252 | 97 (9.6%) | 119 (11.8%) | -0.0712 | 244 (8.0%) | 274 (9.0%) | -0.0359 |
| CV Medication - Mineralocorticoid receptor antagonist ; n (%) CV Medication - Nitrate; n (%) | 573 (44.8%)<br>289 (22.6%) | 578 (45.2%)<br>277 (21.7%) | -0.0080<br>0.0217 | 393 (52.5%)<br>172 (23.0%) | 386 (51.6%)<br>160 (21.4%) | 0.0180 | 443 (44.0%)<br>245 (24.4%) | 427 (42.4%)<br>230 (22.9%) | 0.0323 | 1,016 (33.5%)<br>534 (17.6%) | 1,005 (33.1%)<br>507 (16.7%) | 0.0085 |
| CV Medication - PCSK9 Inhibitors; n (%)* | 0 (0.0%) | 3 (0.2%) | -0.0633 | 2 (0.3%) | 1 (0.1%) | 0.0448 | 3 (0.3%) | 0 (0.0%) | 0.0776 | 003 (0.1%) | 003 (0.1%) | 0.0000 |
| CV Medication - Use of Statins ; n (%) | 907 (70.9%) | 926 (72.4%) | -0.0333 | 495 (66.2%) | 475 (63.5%) | 0.0566 | 728 (72.4%) | 743 (73.9%) | -0.0339 | 1,635 (53.9%) | 1,669 (55.0%) | -0.0221 |
| CV Medication - Use of other lipid-lowering drugs; n (%) CV Medication - CCB (non-dihydropyridine) - Non-combo with ACEi; n (%) | 67 (5.2%)<br>50 (3.9%) | 68 (5.3%)<br>58 (4.5%) | -0.0045<br>-0.0299 | 44 (5.9%)<br>22 (2.9%) | 48 (6.4%)<br>27 (3.6%) | -0.0208<br>-0.0395 | 81 (8.1%)<br>58 (5.8%) | 71 (7.1%)<br>59 (5.9%) | 0.0377<br>-0.0043 | 148 (4.9%)<br>108 (3.6%) | 139 (4.6%)<br>117 (3.9%) | 0.0141<br>-0.0158 |
| CV Medication - CCB (dihydropyridine) - Non-combo with ACEi, ARB; n (%) | 205 (16.0%) | 208 (16.3%) | -0.0082 | 113 (15.1%) | 110 (14.7%) | 0.0112 | 133 (13.2%) | 143 (14.2%) | -0.0291 | 338 (11.1%) | 351 (11.6%) | -0.0158 |
| Other Consolidity Others and (6/) | 60 (4.7%) | 57 (4.5%) | 0.0095 | 21 (2.8%) | 16 (2.1%) | 0.0453 | 74 (7.4%) | 74 (7.40/) | 0.0000 | 134 (4.4%) | 131 (4.3%) | 0.0049 |
| Other Comorbidity - Osteoporosis ; n (%) Other Comorbidity - Dementia ; n (%) | 102 (8.0%) | 57 (4.5%)<br>91 (7.1%) | 0.0095 | 21 (2.8%)<br>36 (4.8%) | 16 (2.1%)<br>36 (4.8%) | 0.0453 | 94 (9.3%) | 74 (7.4%)<br>94 (9.3%) | 0.0000 | 134 (4.4%) | 131 (4.3%) | 0.0049 |
| Other Comorbidity - Hypothyroidism ; n (%) | 40 (3.1%) | 48 (3.8%) | -0.0384 | 28 (3.7%) | 34 (4.5%) | -0.0404 | 76 (7.6%) | 63 (6.3%) | 0.0511 | 116 (3.8%) | 111 (3.7%) | 0.0053 |
| Other Comorbidity - Hyperthyroidism ; n (%) Other Comorbidity - Hyperkalemia ; n (%) | 27 (2.1%)<br>78 (6.1%) | 22 (1.7%)<br>79 (6.2%) | 0.0293<br>-0.0042 | 9 (1.2%)<br>45 (6.0%) | 10 (1.3%)<br>35 (4.7%) | -0.0090<br>0.0578 | 25 (2.5%)<br>70 (7.0%) | 21 (2.1%)<br>68 (6.8%) | 0.0267 | 052 (1.7%)<br>148 (4.9%) | 043 (1.4%)<br>147 (4.8%) | 0.0243<br>0.0047 |
| Other Comorbidity - Pyperkalerina , II (%) Other Comorbidity - Depression; n (%) | 207 (16.2%) | 216 (16.9%) | -0.0042 | 76 (10.2%) | 75 (10.0%) | 0.0066 | 187 (18.6%) | 182 (18.1%) | 0.0129 | 394 (13.0%) | 398 (13.1%) | -0.0030 |
| Other Comorbidity - COPD ; n (%) | 378 (29.6%) | 380 (29.7%) | -0.0022 | 108 (14.4%) | 104 (13.9%) | 0.0143 | 290 (28.8%) | 297 (29.5%) | -0.0154 | 668 (22.0%) | 677 (22.3%) | -0.0072 |
| Other Comorbidity - Pneumonia; n (%) Other Comorbidity - Acute kidney injury (AKI) ; n (%) | 263 (20.6%)<br>284 (22.2%) | 270 (21.1%)<br>321 (25.1%) | -0.0123<br>-0.0683 | 147 (19.7%)<br>158 (21.1%) | 139 (18.6%)<br>150 (20.1%) | 0.0280 | 185 (18.4%)<br>259 (25.7%) | 203 (20.2%)<br>253 (25.1%) | -0.0456<br>0.0138 | 448 (14.8%)<br>543 (17.9%) | 473 (15.6%)<br>574 (18.9%) | -0.0223<br>-0.0258 |
| Other Comorbidity - CKD Stage 1-2; n (%) | 68 (5.3%) | 79 (6.2%) | -0.0387 | 18 (2.4%) | 18 (2.4%) | 0.0000 | 81 (8.1%) | 75 (7.5%) | 0.0224 | 149 (4.9%) | 154 (5.1%) | -0.0092 |
| Other Comorbidity - CKD Stage 3-4; n (%) | 310 (24.2%) | 289 (22.6%) | 0.0378 | 90 (12.0%) | 84 (11.2%) | 0.0250 | 267 (26.5%) | 273 (27.1%) | -0.0135 | 577 (19.0%) | 562 (18.5%) | 0.0128 |
| Other Comorbidity - Any Chronic Kidney Disease; n (%) Other Comorbidity - Hemodialusis (Paritoneal dialusis : n (%) * | 421 (32.9%)<br>7 (0.5%) | 408 (31.9%)<br>4 (0.3%) | 0.0214 | 133 (17.8%) | 125 (16.7%)<br>1 (0.1%) | 0.0291 | 381 (37.9%)<br>4 (0.4%) | 371 (36.9%)<br>0 (0.0%) | 0.0207 | 802 (26.4%)<br>011 (0.4%) | 779 (25.7%)<br>004 (0.1%) | 0.0159 |
| Other Comorbidity - Hemodialysis/Peritoneal dialysis ; n (%)* Other Comorbidity - DM Related Complications; n (%) | 289 (22.6%) | 304 (23.8%) | -0.0284 | 118 (15.8%) | 115 (15.4%) | 0.0000 | 235 (23.4%) | 224 (22.3%) | 0.0896 | 524 (17.3%) | 528 (17.4%) | -0.0026 |
| Other Comorbidity - Diabetic/Hypertensive Nephropathy; n (%) | 419 (32.8%) | 402 (31.4%) | 0.0300 | 143 (19.1%) | 141 (18.9%) | 0.0051 | 329 (32.7%) | 319 (31.7%) | 0.0214 | 748 (24.7%) | 721 (23.8%) | 0.0210 |
| Other Comorbidity - Sleep apnea; n (%) Other Comorbidity - Cancer; n (%) | 298 (23.3%)<br>150 (11.7%) | 307 (24.0%)<br>150 (11.7%) | -0.0165<br>0.0000 | 171 (22.9%)<br>58 (7.8%) | 177 (23.7%)<br>56 (7.5%) | -0.0189<br>0.0113 | 177 (17.6%)<br>126 (12.5%) | 189 (18.8%)<br>131 (13.0%) | -0.0311<br>-0.0150 | 475 (15.7%)<br>276 (9.1%) | 496 (16.4%)<br>281 (9.3%) | -0.0191<br>-0.0069 |
| Other Comorbidity - Type 1 DM ; n (%) | 40 (3.1%) | 47 (3.7%) | -0.0331 | 24 (3.2%) | 22 (2.9%) | 0.0113 | 36 (3.6%) | 40 (4.0%) | -0.0130 | 076 (2.5%) | 087 (2.9%) | -0.0247 |
| Other Comorbidity - Type 2 DM ; n (%) | 662 (51.8%) | 673 (52.6%) | -0.0160 | 348 (46.5%) | 322 (43.0%) | 0.0704 | 531 (52.8%) | 504 (50.1%) | 0.0540 | 1,193 (39.3%) | 1,177 (38.8%) | 0.0102 |
| Other Comorbidity - Anemia ; n (%) | 380 (29.7%) | 356 (27.8%) | 0.0420 | 155 (20.7%) | 144 (19.3%) | 0.0350 | 340 (33.8%) | 348 (34.6%) | -0.0169 | 720 (23.7%) | 704 (23.2%) | 0.0118 |
| Lifestyle - Obesity ; n (%) | 407 (31.8%) | 437 (34.2%) | -0.0511 | 222 (29.7%) | 222 (29.7%) | 0.0000 | 236 (23.5%) | 239 (23.8%) | -0.0071 | 643 (21.2%) | 676 (22.3%) | -0.0267 |
| Lifestyle - Alcohol/Drug Abuse or Dependence; n (%) | 113 (8.8%) | 122 (9.5%) | -0.0243 | 66 (8.8%) | 64 (8.6%) | 0.0071 | 60 (6.0%) | 56 (5.6%) | 0.0171 | 173 (5.7%) | 178 (5.9%) | -0.0086 |
| Lifestyle - Smoking; n (%) | 613 (47.9%) | 628 (49.1%) | -0.0240 | 181 (24.2%) | 163 (21.8%) | 0.0571 | 440 (43.7%) | 436 (43.3%) | 0.0081 | 1,053 (34.7%) | 1,064 (35.1%) | -0.0084 |
| | | 4 (0.3%) | 0.0169 | 5 (0.7%) | 2 (0.3%) | 0.0567 | 11 (1.1%) | 7 (0.7%) | 0.0424 | 016 (0.5%) | 011 (0.4%) | 0.0149 |
| Other Medication - AGI & Meglitinides ; n (%)* | 5 (0.4%) | | | 3 (0.7%) | | | | | | | | |
| Other Medication - AGI & Meglitinides ; n (%)* Other Medication - Insulin; n (%) Other Medication - Gittazones; n (%) | 5 (0.4%)<br>192 (15.0%)<br>17 (1.3%) | 210 (16.4%)<br>20 (1.6%) | -0.0385<br>-0.0251 | 129 (17.2%)<br>15 (2.0%) | 108 (14.4%)<br>11 (1.5%) | 0.0768 | 162 (16.1%)<br>17 (1.7%) | 150 (14.9%)<br>18 (1.8%) | 0.0332 | 354 (11.7%)<br>034 (1.1%) | 360 (11.9%)<br>038 (1.3%) | -0.0062<br>-0.0184 |

| Other Madicalian DDD 4 Inhibitant in (6/) | 00 (7.0%) | 85 (6.6%) | 0.0159 | FC (7 F0/) | 46 (6.1%) | 0.0556 | 00 (0 00/) | 85 (8.4%) | 0.0470 | 400 (5.00/) | 170 (5.6%) | 0.0129 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Other Medication - DPP-4 Inhibitors ; n (%) Other Medication - GLP-1 RA ; n (%) | 90 (7.0%)<br>51 (4.0%) | 85 (6.6%)<br>51 (4.0%) | 0.0159 | 56 (7.5%)<br>21 (2.8%) | 46 (6.1%)<br>23 (3.1%) | 0.0556<br>-0.0177 | 90 (8.9%)<br>17 (1.7%) | 85 (8.4%)<br>13 (1.3%) | 0.0178 | 180 (5.9%)<br>068 (2.2%) | 170 (5.6%)<br>064 (2.1%) | 0.0129 |
| Other Medication - GEP-1 RA ; n (%) Other Medication - Metformin : n (%) | 337 (26.3%) | 341 (26.7%) | -0.0091 | 179 (23.9%) | 172 (23.0%) | 0.0212 | 218 (21.7%) | 217 (21.6%) | 0.0329 | 555 (18.3%) | 558 (18.4%) | -0.0026 |
| Other Medication - NSAIDS (COX-2 Selective) ; n (%) | 72 (5.6%) | 64 (5.0%) | 0.0268 | 36 (4.8%) | 31 (4.1%) | 0.0212 | 43 (4.3%) | 43 (4.3%) | 0.0024 | 115 (3.8%) | 107 (3.5%) | 0.0160 |
| Other Medication - NSAIDS (COX-2 Selective) ; n (%) Other Medication - NSAIDS (Non-Selective) ; n (%) | 126 (9.9%) | 129 (10.1%) | -0.0067 | 136 (18.2%) | 137 (18.3%) | -0.0026 | 43 (4.3%)<br>35 (3.5%) | 43 (4.3%)<br>34 (3.4%) | 0.0000 | 161 (5.3%) | 163 (5.4%) | -0.0044 |
| Other Medication - Use of antiplatelet agents : n (%) | 355 (27.8%) | 377 (29.5%) | -0.0376 | 249 (33.3%) | 237 (31.7%) | 0.0342 | 282 (28.0%) | 292 (29.0%) | -0.0222 | 637 (21.0%) | 669 (22.1%) | -0.0268 |
| Other Medication - Use of Antiplatelet agents , If (%) Other Medication - Use of heparin and other low-molecular weight heparins ; n (%)* | 29 (2.3%) | 27 (2.1%) | 0.0136 | 1 (0.1%) | 0 (0.0%) | 0.0342 | 27 (2.7%) | 9 (0.9%) | 0.1357 | 056 (1.8%) | 036 (1.2%) | 0.0268 |
| Other Medication - Use of oral anticoagulants ; n (%) | 478 (37.4%) | 470 (36.7%) | 0.0136 | 255 (34.1%) | 270 (36.1%) | -0.0447 | 429 (42.6%) | 419 (41.7%) | 0.0182 | 907 (29.9%) | 889 (29.3%) | 0.0434 |
| Other Medication - Use of other hypertension drugs; n (%) | 149 (11.6%) | 140 (10.9%) | 0.0222 | 105 (14.0%) | 97 (13.0%) | 0.0293 | 105 (10.4%) | 108 (10.7%) | -0.0098 | 254 (8.4%) | 248 (8.2%) | 0.0072 |
| Other Medication - Use of antipsychotics ; n (%) | 33 (2.6%) | 36 (2.8%) | -0.0123 | 10 (1.3%) | 11 (1.5%) | -0.0170 | 32 (3.2%) | 27 (2.7%) | 0.0296 | 065 (2.1%) | 063 (2.1%) | 0.0000 |
| Other Medication - Use of dementia meds ; n (%) | 35 (2.7%) | 25 (2.0%) | 0.0462 | 15 (2.0%) | 14 (1.9%) | 0.0072 | 33 (3.3%) | 34 (3.4%) | -0.0056 | 068 (2.2%) | 059 (1.9%) | 0.0212 |
| Other Medication - Use of antiparkinsonian meds ; n (%) | 34 (2.7%) | 38 (3.0%) | -0.0180 | 13 (1.7%) | 13 (1.7%) | 0.0072 | 26 (2.6%) | 29 (2.9%) | -0.0036 | 060 (2.2%) | 067 (2.2%) | -0.0139 |
| Other Medication - Use of anxiolytics/hypnotics ; n (%) | 78 (6.1%) | 81 (6.3%) | -0.0180 | 39 (5.2%) | 54 (7.2%) | -0.0830 | 54 (5.4%) | 62 (6.2%) | -0.0342 | 132 (4.4%) | 143 (4.7%) | -0.0139 |
| Other Medication - Use of anticonvulsants ; n (%) | 181 (14.2%) | 194 (15.2%) | -0.0083 | 76 (10.2%) | 68 (9.1%) | 0.0373 | 166 (16.5%) | 165 (16.4%) | 0.0027 | 347 (11.4%) | 359 (11.8%) | -0.0144 |
| Other Medication - Use of anticonvuisants ; n (%) | 306 (23.9%) | 317 (24.8%) | -0.0282 | 159 (21.3%) | 159 (21.3%) | 0.0000 | 284 (28.2%) | 280 (27.8%) | 0.0027 | 590 (19.5%) | 597 (19.7%) | -0.0123 |
| Other Medication - Use of lithium : n (%)* | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 3 (0.4%) | 0 (0.0%) | 0.0896 | 2 (0.2%) | 0 (0.0%) | 0.0633 | 002 (0.1%) | 000 (0.0%) | 0.0447 |
| Other Medication - Use of Benzodiazepine; n (%) | 197 (15.4%) | 187 (14.6%) | 0.0224 | 92 (12.3%) | 104 (13.9%) | -0.0474 | 131 (13.0%) | 141 (14.0%) | -0.0293 | 328 (10.8%) | 328 (10.8%) | 0.0000 |
| Other Medication - Use of opioids ; n (%) | 385 (30.1%) | 386 (30.2%) | -0.0022 | 213 (28.5%) | 206 (27.5%) | 0.0223 | 267 (26.5%) | 281 (27.9%) | -0.0315 | 652 (21.5%) | 667 (22.0%) | -0.0121 |
| Other Medication - Use of COPD/asthma meds ; n (%) | 296 (23.1%) | 269 (21.0%) | 0.0507 | 139 (18.6%) | 152 (20.3%) | -0.0430 | 195 (19.4%) | 218 (21.7%) | -0.0569 | 491 (16.2%) | 487 (16.1%) | 0.0027 |
| Other Medication - Ose or COPD/astrina meds , if (%) | 290 (23.1%) | 209 (21.0%) | 0.0307 | 159 (16.0%) | 132 (20.5%) | -0.0430 | 193 (19.4%) | 210 (21.7%) | -0.0369 | 491 (10.2%) | 467 (10.176) | 0.0027 |
| HU - Bone mineral density; n (%) | 28 (2.2%) | 28 (2.2%) | 0.0000 | 8 (1.1%) | 9 (1.2%) | -0.0094 | 16 (1.6%) | 14 (1.4%) | 0.0165 | 044 (1.5%) | 042 (1.4%) | 0.0084 |
| HU - Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; n (%) | 61 (4.8%) | 55 (4.3%) | 0.0240 | 30 (4.0%) | 27 (3.6%) | 0.0209 | 36 (3.6%) | 41 (4.1%) | -0.0260 | 097 (3.2%) | 096 (3.2%) | 0.0000 |
| HU - Flu vaccine: n (%) | 235 (18.4%) | 238 (18.6%) | -0.0052 | 76 (10.2%) | 83 (11.1%) | -0.0292 | 306 (30.4%) | 304 (30.2%) | 0.0044 | 541 (17.8%) | 542 (17.9%) | -0.0026 |
| HU - Mammogram: n (%) | 63 (4.9%) | 62 (4.8%) | 0.0047 | 36 (4.8%) | 30 (4.0%) | 0.0390 | 51 (5.1%) | 46 (4.6%) | 0.0233 | 114 (3.8%) | 108 (3.6%) | 0.0106 |
| HU - Frailty Score: Empirical Version 365 days | 05 (4.5%) | GE (4.070) | 0.0047 | 30 (4.070) | 50 (4.0%) | 0.0550 | 51 (5.170) | 40 (4.070) | 0.0255 | 114 (5.0%) | 100 (5.070) | 0.0100 |
| mean (sd) | 0.22 (0.06) | 0.22 (0.06) | 0.0000 | 0.20 (0.05) | 0.19 (0.05) | 0.2000 | 0.24 (0.07) | 0.24 (0.07) | 0.0000 | 0.22 (0.06) | 0.22 (0.06) | 0.0000 |
| median [IQR] | 0.21 [0.18, 0.25] | 0.21 [0.18, 0.25] | 0.0000 | 0.18 [0.16, 0.22] | 0.18 [0.16, 0.21] | 0.0000 | 0.22 [0.19, 0.27] | 0.22 [0.19, 0.27] | 0.0000 | 0.21 (0.06) | 0.21 (0.06) | 0.0000 |
| HU - Number of hospitalizations during CAP | 5.22 [5.25/ 5.25] | ciae (ciae) ciae) | | 0.10 (0.10) 0.111 | 5.10 (8.10) 5.111 | | 0.00 (0.00) 0.0. | 0.00 (0.00) 0.00) | | 0.22 (0.00) | (0.00) | |
| mean (sd) | 1.06 (0.77) | 1.08 (0.76) | -0.0261 | 0.98 (0.65) | 0.95 (0.66) | 0.0458 | 1.07 (0.91) | 1.07 (0.90) | 0.0000 | 1.04 (0.79) | 1.04 (0.79) | 0.0000 |
| median [IOR] | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.0000 | 1.00 [1.00, 1.00] | 1.00 [0.75, 1.00] | 0.0000 | 1.00 (0.79) | 1.00 (0.79) | 0.0000 |
| HU - Number of Emergency Department (ED) visits | 2.00 (2.00) 2.00) | 2.00 (2.00) | | () | (2.00) | | () | 200 (00.0) 2000) | | () | 2.00 (0.10) | |
| mean (sd) | 1.81 (2.51) | 1.84 (2.32) | -0.0124 | 2.56 (5.33) | 2.40 (3.90) | 0.0343 | 1.73 (2.19) | 1.65 (2.78) | 0.0320 | 1.97 (3.35) | 1.92 (2.93) | 0.0159 |
| median [IOR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | 0.0000 | 2.00 [0.00, 3.00] | 2.00 [0.00, 3.00] | 0.0000 | 1.00 [0.00, 3.00] | 1.00 [0.00, 2.00] | 0.0000 | 1.25 (3.35) | 1.25 (2.93) | 0.0000 |
| HU - Number of Internal Medicine/Family Medicine Visits | | | | ,, | | | | , | | | | |
| mean (sd) | 14.51 (18.56) | 14.34 (19.30) | 0.0090 | 9.77 (15.50) | 8.91 (12.31) | 0.0614 | 8.50 (9.54) | 8.89 (10.84) | -0.0382 | 11.35 (15.32) | 11.19 (15.28) | 0.0105 |
| median [IOR] | 9.00 [4.00, 18.00] | 9.00 [4.00, 19.00] | 0.0000 | 5.00 [2.00, 11.75] | 5.00 [2.00, 11.00] | 0.0000 | 6.00 [3.00, 11.00] | 6.00 [3.00, 11.00] | 0.0000 | 7.02 (15.32) | 7.02 (15.28) | 0.0000 |
| HU - Number of Distinct Medication Prescriptions (not generalized to generics) | | | | | | | | | | | | |
| mean (sd) | 33.63 (25.85) | 33.96 (20.50) | -0.0141 | 30.49 (17.53) | 30.50 (15.10) | -0.0006 | 31.27 (19.20) | 32.09 (16.13) | -0.0462 | 32.07 (21.91) | 32.49 (17.88) | -0.0210 |
| median [IQR] | 28.00 [19.00, 41.00] | 30.00 [20.00, 43.00] | -0.0857 | 28.00 [19.00, 38.00] | 28.00 [20.00, 38.00] | 0.0000 | 27.00 [19.00, 38.00] | 29.00 [21.00, 40.00] | -0.1128 | 27.67 (21.91) | 29.18 (17.88) | -0.0755 |
| HU - Number of Cardiologist visits | | | | | | | | | | | | |
| mean (sd) | 13.79 (13.06) | 13.37 (10.66) | 0.0352 | 6.17 (8.33) | 6.95 (7.55) | -0.0981 | 11.33 (12.78) | 11.70 (11.61) | -0.0303 | 11.09 (11.97) | 11.23 (10.33) | -0.0125 |
| median [IQR] | 11.00 [5.00, 18.00] | 11.00 [6.00, 18.00] | 0.0000 | 4.00 [0.00, 9.00] | 5.00 [2.00, 10.00] | -0.1258 | 8.00 [3.00, 15.00] | 9.00 [4.00, 15.00] | -0.0819 | 8.28 (11.97) | 8.86 (10.33) | -0.0519 |
| HU - Number of Electrocardiogram | | | | | | | | | | | | |
| mean (sd) | 4.47 (4.88) | 4.32 (4.33) | 0.0325 | 3.27 (3.08) | 3.22 (2.91) | 0.0167 | 3.88 (3.82) | 3.73 (3.96) | 0.0386 | 3.98 (4.15) | 3.85 (3.90) | 0.0323 |
| median [IQR] | 3.00 [1.00, 6.00] | 3.00 [2.00, 6.00] | 0.0000 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0.0000 | 3.00 [1.00, 5.00] | 3.00 [1.00, 5.00] | 0.0000 | 2.75 (4.15) | 2.75 (3.90) | 0.0000 |
| | 5.00 [1.00, 6.00] | | | | 2.00 [1.00, 4.00] | | | | | | | |
| HU - Number of Echocardiogram | 5.00 [1.00, 6.00] | 5.00 [2.00, 0.00] | | | 2.00 [1.00, 4.00] | 0.0000 | | | | | | |
| HU - Number of Echocardiogrammean (sd) | 2.86 (5.89) | 2.82 (5.27) | 0.0072 | 1.78 (2.00) | 1.76 (1.58) | 0.0111 | 1.66 (1.50) | 1.62 (1.34) | 0.0281 | 2.20 (4.05) | 2.16 (3.60) | 0.0104 |
| | | | | | | | | 1.62 (1.34)<br>1.00 [1.00, 2.00] | 0.0281<br>0.0000 | 2.20 (4.05)<br>1.00 (4.05) | 2.16 (3.60)<br>1.00 (3.60) | 0.0104<br>0.0000 |
| mean (sd) | 2.86 (5.89) | 2.82 (5.27) | 0.0072 | 1.78 (2.00) | 1.76 (1.58) | 0.0111 | 1.66 (1.50) | | | | | |
| mean (sd)median [IQR] | 2.86 (5.89) | 2.82 (5.27) | 0.0072 | 1.78 (2.00) | 1.76 (1.58) | 0.0111 | 1.66 (1.50) | | | | | |
| mean (sd)median [lQR] SES Prow - Copay for pharmacy cost (charges in U.S. 5) | 2.86 (5.89)<br>1.00 [1.00, 3.00] | 2.82 (5.27)<br>1.00 [1.00, 3.00] | 0.0072<br>0.0000<br>0.0359<br>-0.0600 | 1.78 (2.00)<br>1.00 [1.00, 2.00] | 1.76 (1.58)<br>1.00 [1.00, 2.00] | 0.0111<br>0.0000<br>0.0074<br>-0.1150 | 1.66 (1.50)<br>1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | -0.0000<br>-0.0053<br>-0.0796 | 1.00 (4.05) | 1.00 (3.60) | 0.0000<br>0.0167<br>-0.0719 |
| mean (sd)median IQR SES Proxy - Copay for pharmacy cost (charges in U.S. \$)mean (sd) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41) | 0.0072<br>0.0000<br>0.0359 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 (14.06) | 0.0111<br>0.0000<br>0.0074 | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56) | 1.00 [1.00, 2.00]<br>26.03 (30.53) | -0.0053 | 1.00 (4.05)<br>23.71 (36.11) | 1.00 (3.60)<br>23.18 (26.88) | 0.0000 |
| median [IQR] SES Proxy - Copay for pharmacy cost (charges in U.S. S)mean [sd]median [IQR] | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88] | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73] | 0.0072<br>0.0000<br>0.0359<br>-0.0600 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38] | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 (14.06)<br>12.40 [5.11, 19.94] | 0.0111<br>0.0000<br>0.0074<br>-0.1150 | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03] | 1.00 [1.00, 2.00]<br>26.03 (30.53)<br>18.78 [5.57, 34.95] | -0.0000<br>-0.0053<br>-0.0796 | 1.00 (4.05)<br>23.71 (36.11)<br>14.65 (36.11) | 1.00 (3.60)<br>23.18 (26.88)<br>16.94 (26.88) | 0.0000<br>0.0167<br>-0.0719 |
| mean (sd)median [QR] SES Proxy - Copay for pharmacy cost (charges in U.S. 5)mean (sd)median [QR] SES Proxy - Low income indicator; n (%) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 (21.5%)<br>325 (25.4%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 (6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 [14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150 | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%) | 1.00 [1.00, 2.00]<br>26.03 (30.53)<br>18.78 [5.57, 34.95]<br>0 (0.0%) | 0.0000<br>-0.0053<br>-0.0796<br>#DIV/0! | 1.00 (4.05)<br>23.71 (36.11)<br>14.65 (36.11)<br>275 (9.1%)<br>325 (10.7%) | 1.00 (3.60)<br>23.18 (26.88)<br>16.94 (26.88) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273 |
| medan [GR] SES Proxy - Copay for pharmacy cost (charges in U.S. 5)mean [GR]median [IQR] SES Proxy - Low income indicator; n (%) SES Proxy - Low income indicator; n (%) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 (21.5%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73]<br>299 (23.4%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 (14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0! | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%) | 1.00 [1.00, 2.00]<br>26.03 (30.53)<br>18.78 [5.57, 34.95]<br>0 (0.0%) | 0.0000<br>-0.0053<br>-0.0796<br>#DIV/0! | 1.00 (4.05)<br>23.71 (36.11)<br>14.65 (36.11)<br>275 (9.1%) | 1.00 (3.60)<br>23.18 (26.88)<br>16.94 (26.88)<br>299 (9.9%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273 |
| median [IQR] SES Proxy - Copay for pharmacy cost (charges in U.S. \$)mean [sd]median [IQR] SES Proxy - Low income indicator; n (%) SES Proxy - Business typecommercial; n (%) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 (21.5%)<br>325 (25.4%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%)<br>939 (73.4%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 [14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%)<br>0 (0.0%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0! | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%) | 1.00 [1.00, 2.00] 26.03 (30.53) 18.78 [5.57, 34.95] 0 (0.0%) 0 (0.0%) | 0.0000<br>-0.0053<br>-0.0796<br>#DIV/0! | 1.00 (4.05)<br>23.71 (36.11)<br>14.65 (36.11)<br>275 (9.1%)<br>325 (10.7%) | 1.00 (3.60)<br>23.18 (26.88)<br>16.94 (26.88)<br>299 (9.9%)<br>340 (11.2%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273<br>-0.0160<br>0.0108 |
| median (IQR) SES Proxy - Copay for pharmacy cost (charges in U.S. 5)median (IQR)median (IQR) SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%)Medicare, n (%) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 (21.5%)<br>325 (25.4%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 (6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 [14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0!<br>#DIV/0!<br>#DIV/0! | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%) | 1.00 [1.00, 2.00]<br>26.03 (30.53)<br>18.78 [5.57, 34.95]<br>0 (0.0%) | 0.0000<br>-0.0053<br>-0.0796<br>#DIV/0! | 1.00 (4.05)<br>23.71 (36.11)<br>14.65 (36.11)<br>275 (9.1%)<br>325 (10.7%) | 1.00 (3.60)<br>23.18 (26.88)<br>16.94 (26.88)<br>299 (9.9%)<br>340 (11.2%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273 |
| median [IQR] SES Proxy - Copay for pharmacy cost (charges in U.S. \$)mean [sd]median [IQR] SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%)Medicare; n (%) SES Proxy - Business type | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 [21.5%]<br>325 (25.4%)<br>954 (74.6%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%)<br>939 (73.4%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455<br>-0.0274 | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%)<br>0 (0.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 [14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%)<br>0 (0.0%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0!<br>#DIV/0! | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%)<br>0 (0.0%) | 1.00 [1.00, 2.00] 26.03 (30.53) 18.78 [5.57, 34.95] 0 (0.0%) 0 (0.0%) | 0.0000 -0.0053 -0.0796 #DIV/0! #DIV/0! | 1.00 (4.05) 23.71 (36.11) 14.65 (36.11) 275 (9.1%) 325 (10.7%) 954 (31.5%) | 1.00 (3.60) 23.18 (26.88) 16.94 (26.88) 299 (9.9%) 340 (11.2%) 939 (31.0%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273<br>-0.0160<br>0.0108 |
| median (IQR) SES Proxy - Copay for pharmacy cost (charges in U.S. 5)median (IQR)median (IQR) SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%)Medicare; n (%) SES Proxy - Insurance Plan typeComprehensive; n (%) | 2.86 (5.89)<br>1.00 [1.00, 3.00]<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 [21.5%]<br>325 [25.4%]<br>954 [74.6%]<br>0 (0.0%)<br>0 (0.0%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%)<br>339 (73.4%)<br>0 (0.0%)<br>0 (0.0%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455<br>-0.0274<br>0.0274<br>#DIV/0!<br>#DIV/0! | 1.78 (2.00)<br>1.00 [1.00, 2.00]<br>14.87 (18.19)<br>10.53 [3.58, 20.38]<br>0 (0.0%)<br>0 (0.0%)<br>105 (14.0%) | 1.76 (1.58)<br>1.00 [1.00, 2.00]<br>14.75 (14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%)<br>0 (0.0%)<br>94 (12.6%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.0412<br>-0.0422<br>0.0080 | 1.66 (1.50) 1.00 [1.00, 2.00] 25.85 (36.56) 16.10 [5.26, 32.03] 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 1.00 [1.00, 2.00] 26.03 (30.53) 18.78 [5.57, 34.95] 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 0.0000 -0.0053 -0.0796 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/O! #DIV/O! #DIV/O! | 1.00 (4.05) 23.71 (36.11) 14.65 (36.11) 275 (9.1%) 325 (10.7%) 954 (31.5%) 105 (3.5%) | 1.00 (3.60) 23.18 (26.88) 16.94 (26.88) 299 (9.9%) 340 (11.2%) 939 (31.0%) 094 (3.1%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273<br>-0.0160<br>0.0108<br>-0.0224<br>-0.0207<br>0.0029 |
| median [IQR] SES Proxy - Copay for pharmacy cost (charges in U.S. S)mean [sd]median [IQR] SES Proxy - Low income indicator; n (%) SES Proxy - Business typeCommercial; n (%)Medicare; n (%)Medicare; n (%) SES Proxy - Business StypeCommercial; n (%)Medicare; n (%)Medicare; n (%) | 2.86 (5.89)<br>1.00 (1.00, 3.00)<br>27.20 (42.97)<br>15.93 [5.74, 32.88]<br>275 (212.5%)<br>325 (25.4%)<br>954 (74.6%)<br>0 (0.0%)<br>0 (0.0%) | 2.82 (5.27)<br>1.00 [1.00, 3.00]<br>25.88 (29.41)<br>18.14 [6.52, 33.73]<br>299 (23.4%)<br>340 (26.6%)<br>939 (73.4%)<br>0 (0.0%)<br>0 (0.0%) | 0.0072<br>0.0000<br>0.0359<br>-0.0600<br>-0.0455<br>-0.0274<br>0.0274<br>#DIV/0! | 1.78 (2.00)<br>1.00 (1.00, 2.00)<br>14.87 (18.19)<br>10.53 (3.58, 20.38)<br>0 (0.0%)<br>0 (0.0%)<br>105 (14.0%)<br>62 (8.3%) | 1.76 (1.58)<br>1.00 (1.00, 2.00)<br>14.75 (14.06)<br>12.40 [5.11, 19.94]<br>0 (0.0%)<br>0 (0.0%)<br>94 (12.6%)<br>71 (9.5%) | 0.0111<br>0.0000<br>0.0074<br>-0.1150<br>#DIV/0!<br>#DIV/0!<br>#DIV/0!<br>0.0412<br>-0.0422 | 1.66 (1.50)<br>1.00 [1.00, 2.00]<br>25.85 (36.56)<br>16.10 [5.26, 32.03]<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%)<br>0 (0.0%) | 1.00 [1.00, 2.00] 26.03 (30.53) 18.78 [5.57, 34.95] 0 (0.0%) 0 (0.0%) 0 (0.0%) 0 (0.0%) | 0.0000 -0.0053 -0.0796 #DIV/0! #DIV/0! #DIV/0! #DIV/0! #DIV/0! | 1.00 (4.05) 23.71 (36.11) 14.65 (36.11) 275 (9.1%) 325 (10.7%) 954 (31.5%) 105 (3.5%) 062 (2.0%) | 1.00 (3.60) 23.18 (26.88) 16.94 (26.88) 299 (9.9%) 340 (11.2%) 939 (31.0%) 094 (3.1%) 071 (2.3%) | 0.0000<br>0.0167<br>-0.0719<br>-0.0273<br>-0.0160<br>0.0108<br>0.0224<br>-0.0207 |

<sup>\*</sup>Excluded from PS model: Age Cateogries, Use of Lithium, Use of AGI & Meglinitides, PCSK9 Inhibitors, Use of heparin or LMWH, Hemodialysis/Peritoneal dialysis